CLINICAL TRIAL: NCT02912650
Title: A Phase 3, Double-Blind, Randomized, Safety And Efficacy Study Comparing A Single Oral Dose Of Ibuprofen (IBU) 250 Mg/Acetaminophen (APAP) 500 Mg (Administered As Two Tablets Of IBU/APAP 125 Mg/250 Mg) To Each Active Drug Monocomponent Alone And To Placebo In The Treatment Of Post-Surgical Dental Pain
Brief Title: A Safety And Efficacy Study of Ibuprofen 250 mg / Acetaminophen 500 mg In The Treatment Of Post-Surgical Dental Pain
Acronym: SDDP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B5061003; GEMINI SDDP (Other: Alias Study Number)
Record Dates: First submitted 2016-01-07; First posted 2016-09-23 (Estimated); Results first posted 2017-08-30 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-07

CONDITIONS: Post-surgical Pain Following Extraction of Molar Teeth
Keywords: ibuprofen; acetaminophen; pain; molar extraction
MeSH Terms: conditions — Pain | interventions — Ibuprofen; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ibuprofen 250 mg / Acetaminophen 500 mg (Experimental): 2 caplets of Ibuprofen 125 mg / Acetaminophen 250 mg
  Interventions: Drug: Ibuprofen 250 mg / Acetaminophen 500 mg
- Ibuprofen 250 mg (Active Comparator): 2 caplets of IBU 125 mg
  Interventions: Drug: Ibuprofen 250 mg
- Acetaminophen 650 mg (Active Comparator): 2 tablets of APAP 325 mg
  Interventions: Drug: Acetaminophen 650 mg
- Placebo (Active Comparator): 2 caplets of Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ibuprofen 250 mg / Acetaminophen 500 mg — 2 caplets of Ibuprofen 250 mg / Acetaminophen 500 mg
  Other Names: IBU 250 / APAP 500
  Arms: Ibuprofen 250 mg / Acetaminophen 500 mg
Drug: Ibuprofen 250 mg — 2 caplets of Ibuprofen 125 mg
  Other Names: IBU 250
  Arms: Ibuprofen 250 mg
Drug: Acetaminophen 650 mg — 2 tablets of Acetaminophen 325 mg
  Other Names: APAP 650
  Arms: Acetaminophen 650 mg
Drug: Placebo — 2 caplets of Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double blind, placebo-controlled, parallel group, single-center study in approximately 560 subjects to determine the overall analgesic efficacy and safety of a fixed-dose ibuprofen 250 mg / acetaminophen 500 mg formulation compared to ibuprofen 250 mg alone, acetaminophen 650 mg alone, and to placebo. Subjects will be healthy males and females aged 18-40 years, inclusive, who are experiencing post-operative pain following surgical extraction of 3 or more third molar teeth. Following extraction, subjects must experience, within 5 hours, post-surgical pain of at least moderate severity (on a 4-point categorical scale), confirmed by a Visual Analog Pain Severity Rating Scale (VAS PSR) of at least 50 mm on a 100 mm VAS PSR scale. Eligible subjects will be randomized to receive a single oral dose of study medication under double-blind conditions and then evaluated on site for 12 hours following administration of study medication. Subjects will provide self-ratings of pain severity and pain relief at various time points using categorical and numerical scales. Additionally, subjects will also evaluate the time to first perceptible relief and time to meaningful relief using a double stopwatch method. Finally, at 12 hours, subjects will complete a categorical Global Evaluation of the study medication. A review of any reported adverse events will also be completed.

DETAILED DESCRIPTION:
This is a 12-hour, 4-arm, randomized, double blind, placebo-controlled, parallel group, single-center study in approximately 560 subjects to determine the overall analgesic efficacy and safety of a fixed-dose ibuprofen 250 mg / acetaminophen 500 mg formulation (administered as two caplets of 125 mg/250 mg IBU/APAP) compared to ibuprofen 250 mg alone, acetaminophen 650 mg alone, and to placebo. Subjects will be healthy males and females aged 18-40 years, inclusive, otherwise healthy, who are experiencing post-operative pain following surgical extraction of 3 or more third molar teeth. Following extraction, subjects must experience, within 5 hours, post-surgical pain of at least moderate severity (on a 4-point categorical scale), confirmed by a Visual Analog Pain Severity Rating Scale (VAS PSR) of at least 50 mm on a 100 mm VAS PSR scale. Upon completion of the baseline scales, eligible subjects will be randomized to receive a single oral dose of study medication under double-blind conditions and then evaluated on site for 12 hours following administration of study medication. At 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12 hours post dose time points, subjects will provide: self-ratings of pain severity using the numerical and categorical PSRs; and self-ratings of pain relief at each time point using a categorical pain relief rating scale. At 12 hours, subjects will also complete a 6-point categorical Global Evaluation of the study medication. Additionally, subjects will also evaluate the time to first perceptible relief and time to meaningful relief using a double stopwatch method up to 12 hours post-dose or until the time of first rescue medication use, whichever is sooner. A review of any reported adverse events will also be completed.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients who have undergone surgical extraction of 3 or more third molars, of which at least 2 must be a partial or complete bony mandibular impaction.
* Subject must have at least moderate pain on the 4-point categorical scale, confirmed by at least 50 mm on the 100 mm VAS PSR scale within approximately 5 hours (i.e., less than or equal to 5 hours, 15 minutes) after surgery is completed.
* Female subjects are not pregnant or breast feeding.
* Informed consent.

Exclusion Criteria:

* Presence or history of any significant hepatic, renal, endocrine, cardiovascular, neurological, psychiatric, gastrointestinal, pulmonary, hematologic, or metabolic disorder determined by the Investigator to place the subject at increased risk, including the presence or history within 2 years of screening.
* Acute localized dental alveolar infection at the time of surgery that could confound the post-surgical evaluation.
* Hypersensitivity to ibuprofen, naproxen, aspirin, or any other NSAID; or to APAP, tramadol, other opioids, or to their combinations.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 568 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Jean Brown Research, Salt Lake City, Utah, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B5061003&StudyName=A%20Phase%203%2C%20Double-blind%2C%20Randomized%2C%20Safety%20And%20Efficacy%20Study%20Comparing%20A%20Single%20Oral%20Dose%20Of%20Ibuprofen%20%28ibu%29%20250%20Mg%2Facetaminophen%20%28apap%29%20500%20Mg%20%28administered%20As%20Two%20Tablets%20Of%20Ibu%2Fapap%20125%20Mg%2F250%20Mg%29%20To%20Each%20Active%20Drug%20Monocomponent%20Alone%20And%20To%20Placebo%20In%20The%20Treatment%20Of%20Post-surgical%20Dental%20Pain

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received Placebo as a single oral dose caplet during the study of 12 hours.
- Ibuprofen 250 mg + Acetaminophen 500 mg: Participants received a single oral dose of a fixed dose combination of ibuprofen 250 milligram (mg) and acetaminophen 500 mg caplets during the 12 hours study.
- Ibuprofen 250 mg: Participants received a single oral dose of ibuprofen 250 mg caplet, during the 12 hours study.
- Acetaminophen 650 mg: Participants received a single oral dose of acetaminophen 650 mg tablet, during the 12 hours study.
Period: Overall Study
Arm/Group | Placebo | Ibuprofen 250 mg + Acetaminophen 500 mg | Ibuprofen 250 mg | Acetaminophen 650 mg
Started | 56 | 172 | 175 | 165
Completed | 55 | 172 | 173 | 160
Not Completed | 1 | 0 | 2 | 5
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 5
Not completed — Adverse Event | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized participants who were dosed with the study medication and provided a baseline assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ibuprofen 250 mg + Acetaminophen 500 mg | Ibuprofen 250 mg | Acetaminophen 650 mg | Total
Number analyzed (Participants) | 56 | 172 | 175 | 165 | 568
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.6 (3.0) | 19.3 (1.8) | 19.7 (2.7) | 19.4 (2.1) | 19.5 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 102 | 102 | 97 | 335
  Male | 22 | 70 | 73 | 68 | 233

OUTCOME MEASURES:

1. Primary Outcome: Time-weighted Sum of Pain Intensity Difference Scores on 11-Point Numerical Scale From 0 to 8 Hours Post-dose (SPID11 [0-8])
Description: Pain intensity was assessed on an 11-point numerical pain severity rating scale. SPID11 (0-8): Time-weighted sum of pain intensity difference (PID) scores over 8 hours. SPID11 score range was -40 (worst score) to 80 (best score) for SPID 0-8. PID was calculated by subtracting the pain intensity score at given post-dose time points (pain severity score range: 0 =no pain to 10 =worst possible pain) from the baseline pain intensity scores (score range: 5 =moderate pain to 10 =worst possible pain; as participants with baseline pain score of at least moderate were included in study). Total possible score range for PID: -5 (worst score) to 10 (best score).
Time Frame: 0 to 8 hours post-dose
Population: FAS included all randomized participants who were dosed with the study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen 250 mg + Acetaminophen 500 mg | Ibuprofen 250 mg | Acetaminophen 650 mg
Number analyzed (Participants) | 56 | 172 | 175 | 165
units on a scale | 4.1 (19.0) | 34.3 (19.6) | 28.9 (20.5) | 19.4 (20.0)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; Treatment difference and 95 percent (%) confidence interval (CI) were based on LS Mean from analysis of covariance (ANCOVA) with treatment, gender, baseline categorical pain severity rating (PSR) as classification variables and baseline numerical PSR used as a continuous covariate; Test type: Superiority or Other; p < 0.001, ANCOVA; Least Squares (LS) Mean Difference = 30.08, 95% CI 2-sided [24.14 to 36.02]
Statistical Analysis 2: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; Treatment difference and 95% CI were based on LS Mean from ANCOVA with treatment, gender, baseline categorical PSR as classification variables and baseline numerical PSR used as a continuous covariate; Test type: Superiority or Other; p = 0.008, ANCOVA; LS Mean Difference = 5.66, 95% CI 2-sided [1.51 to 9.80]
Statistical Analysis 3: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 14.76, 95% CI 2-sided [10.55 to 18.97]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 24.42, 95% CI 2-sided [18.50 to 30.35]
Statistical Analysis 5: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 15.32, 95% CI 2-sided [9.35 to 21.29]
Statistical Analysis 6: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 9.10, 95% CI 2-sided [4.90 to 13.31]

2. Secondary Outcome: Time-weighted Sum of Pain Intensity Difference Scores on 11-Point Numerical Scale From 6 to 8 Hours Post-dose (SPID11 [6-8])
Description: Pain intensity was assessed on an 11-point numerical pain severity rating scale. SPID11 (6-8): Time-weighted sum of PID scores over 6 to 8 hours. SPID11 score range was -15 (worst score) to 30 (best score) for SPID 6-8. PID was calculated by subtracting the pain intensity score at given post-dose time points (pain severity score range: 0 =no pain to 10 =worst possible pain) from the baseline pain intensity scores (score range: 5 =moderate pain to 10 =worst possible pain; as participants with baseline pain score of at least moderate were included in study). Total possible score range for PID: -5 (worst score) to 10 (best score).
Time Frame: 6 to 8 hours post-dose
Population: FAS included all randomized participants who were dosed with the study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen 250 mg + Acetaminophen 500 mg | Ibuprofen 250 mg | Acetaminophen 650 mg
Number analyzed (Participants) | 56 | 172 | 175 | 165
units on a scale | 1.9 (8.8) | 11.3 (9.2) | 9.5 (8.9) | 5.6 (8.8)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 9.26, 95% CI 2-sided [6.59 to 11.94]
Statistical Analysis 2: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.053, ANCOVA; LS Mean Difference = 1.84, 95% CI 2-sided [-0.03 to 3.71]
Statistical Analysis 3: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 5.59, 95% CI 2-sided [3.69 to 7.49]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 7.42, 95% CI 2-sided [4.75 to 10.09]
Statistical Analysis 5: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.008, ANCOVA; LS Mean Difference = 3.67, 95% CI 2-sided [0.98 to 6.36]
Statistical Analysis 6: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 3.75, 95% CI 2-sided [1.85 to 5.64]

3. Secondary Outcome: Time-weighted Sum of Pain Relief Rating (TOTPAR) From 0 to 8 Hours and 6 to 8 Hours Post-dose
Description: TOTPAR: Time-weighted sum of Pain Relief Rating (PRR) scores over 0 to 8 and 6 to 8 hours. TOTPAR total score range: 0 (worst score) to 32 (best score) for TOTPAR 0-8 and 0 (worst score) to 12 (best score) for TOTPAR 6-8 hours. PRR was assessed on a 5-point categorical pain relief rating scale which ranges from 0 =no relief to 4 =complete relief.
Time Frame: 0 to 8 hours, 6 to 8 hours post-dose
Population: FAS included all randomized participants who were dosed with the study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen 250 mg + Acetaminophen 500 mg | Ibuprofen 250 mg | Acetaminophen 650 mg
Number analyzed (Participants) | 56 | 172 | 175 | 165
units on a scale
  0 to 8 hours | 5.3 (7.9) | 18.4 (8.5) | 15.4 (9.0) | 11.4 (9.1)
  6 to 8 hours | 2.3 (3.8) | 6.2 (4.1) | 5.1 (4.0) | 3.5 (4.0)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 0-8 hours: Treatment difference and 95% CI were based on LS Mean from analysis of variance (ANOVA) with treatment, gender and baseline categorical PSR; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 13.05, 95% CI 2-sided [10.39 to 15.71]
Statistical Analysis 2: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; 0 to 8 hours: Treatment difference and 95% CI were based on LS Mean from ANOVA with treatment, gender and baseline categorical PSR; Test type: Superiority or Other; p = 0.002, ANOVA; LS Mean Difference = 3.01, 95% CI 2-sided [1.15 to 4.86]
Statistical Analysis 3: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 6.94, 95% CI 2-sided [5.06 to 8.83]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 10.05, 95% CI 2-sided [7.39 to 12.70]
Statistical Analysis 5: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 6.11, 95% CI 2-sided [3.44 to 8.78]
Statistical Analysis 6: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 3.94, 95% CI 2-sided [2.06 to 5.81]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 6 to 8 hours: Treatment difference and 95% CI were based on LS Mean from ANOVA with treatment, gender and baseline categorical PSR; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 3.84, 95% CI 2-sided [2.63 to 5.05]
Statistical Analysis 8: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 3, analysis 7]; Test type: Superiority or Other; p = 0.013, ANOVA; LS Mean Difference = 1.07, 95% CI 2-sided [0.23 to 1.92]
Statistical Analysis 9: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 3, analysis 7]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 2.69, 95% CI 2-sided [1.83 to 3.55]
Statistical Analysis 10: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 3, analysis 7]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 2.77, 95% CI 2-sided [1.56 to 3.98]
Statistical Analysis 11: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 3, analysis 7]; Test type: Superiority or Other; p = 0.064, ANOVA; LS Mean Difference = 1.15, 95% CI 2-sided [-0.07 to 2.37]
Statistical Analysis 12: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 3, analysis 7]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.62, 95% CI 2-sided [0.76 to 2.47]

4. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure was defined as the time interval from the study drug administration up to the first documentation of treatment failure. Treatment failure was defined as taking the rescue medication or discontinuation of the participants from the study due to lack of efficacy, whichever came first. Participants were censored at 12 hours or at their final assessment time, whichever came first.
Time Frame: 0 to 12 hours post-dose
Population: FAS included all randomized participants who were dosed with the study medication and provided a baseline assessment.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Ibuprofen 250 mg + Acetaminophen 500 mg | Ibuprofen 250 mg | Acetaminophen 650 mg
Number analyzed (Participants) | 56 | 172 | 175 | 165
minutes | 107.0 (8.8) [86.0 to 173.0] | 629.0 (9.2) [570.0 to 720.0] | 608.5 (8.9) [545.0 to 671.0] | 449.0 (8.8) [399.0 to 547.0]
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; p-value was calculated by using Gehan-Wilcoxon test, stratified by gender and baseline categorical PSR terms; Test type: Superiority or Other; p < 0.001, Gehan-Wilcoxon test
Statistical Analysis 2: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; p-value was calculated by using Gehan-Wilcoxon test, stratified by gender and baseline categorical PSR terms; Test type: Superiority or Other; p = 0.069, Gehan-Wilcoxon test
Statistical Analysis 3: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; p-value was calculated by using Gehan-Wilcoxon test, stratified by gender and baseline categorical PSR terms; Test type: Superiority or Other; p < 0.001, Gehan-Wilcoxon test
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen 250 mg; p-value was calculated by using Gehan-Wilcoxon test, stratified by gender and baseline categorical PSR terms; Test type: Superiority or Other; p < 0.001, Gehan-Wilcoxon test
Statistical Analysis 5: Comparison: Placebo vs Acetaminophen 650 mg; p-value was calculated by using Gehan-Wilcoxon test, stratified by gender and baseline categorical PSR terms; Test type: Superiority or Other; p < 0.001, Gehan-Wilcoxon test
Statistical Analysis 6: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; p-value was calculated by using Gehan-Wilcoxon test, stratified by gender and baseline categorical PSR terms; Test type: Superiority or Other; p = 0.005, Gehan-Wilcoxon test

5. Secondary Outcome: Cumulative Percentage of Participants With Treatment Failure at 6 and 8 Hours
Description: Treatment failure was defined as taking the rescue medication or discontinuation of the participants from the study due to lack of efficacy, whichever came first. Participants were censored at 12 hours or at their final assessment time, whichever came first. Percentage of participants who had treatment failure were reported.
Time Frame: 6 hours, 8 hours post-dose
Population: FAS included all randomized participants who were dosed with the study medication and provided a baseline assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ibuprofen 250 mg + Acetaminophen 500 mg | Ibuprofen 250 mg | Acetaminophen 650 mg
Number analyzed (Participants) | 56 | 172 | 175 | 165
percentage of participants
  6 hour | 67.9 (7.9) | 10.5 (8.5) | 21.7 (9.0) | 38.8 (9.1)
  8 hour | 69.6 (3.8) | 24.4 (4.1) | 33.1 (4.0) | 51.5 (4.0)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; At 8 hour: Treatment difference and its associated 95% CI were calculated based on Cochran-Mantel-Haenszel (CMH) adjusted proportions, controlling for baseline categorical PSR and gender using table scores; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -45.27, 95% CI 2-sided [-58.96 to -31.58]
Statistical Analysis 2: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; At 8 hour: Treatment difference and its associated 95% CI were calculated based on CMH adjusted proportions, controlling for baseline categorical PSR and gender using table scores; Test type: Superiority or Other; p = 0.064, Cochran-Mantel-Haenszel; CMH adjusted proportions = -8.88, 95% CI 2-sided [-18.27 to 0.50]
Statistical Analysis 3: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p < 0.001, ANOVA; CMH adjusted proportions = -26.98, 95% CI 2-sided [-36.91 to -17.05]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -36.26, 95% CI 2-sided [-50.45 to -22.07]
Statistical Analysis 5: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p = 0.010, Cochran-Mantel-Haenszel; CMH adjusted proportions = -18.58, 95% CI 2-sided [-32.64 to -4.52]
Statistical Analysis 6: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -18.17, 95% CI 2-sided [-28.44 to -7.90]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; At 6 hour: Treatment difference and its associated 95% CI were calculated based on CMH adjusted proportions, controlling for baseline categorical PSR and gender using table scores; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -57.58, 95% CI 2-sided [-70.44 to -44.72]
Statistical Analysis 8: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; p = 0.004, Cochran-Mantel-Haenszel; CMH adjusted proportions = -11.28, 95% CI 2-sided [-18.99 to -3.57]
Statistical Analysis 9: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -28.06, 95% CI 2-sided [-36.77 to -19.35]
Statistical Analysis 10: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -46.01, 95% CI 2-sided [-59.98 to -32.04]
Statistical Analysis 11: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -29.70, 95% CI 2-sided [-43.65 to -15.75]
Statistical Analysis 12: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -16.94, 95% CI 2-sided [-26.59 to -7.29]

6. Secondary Outcome: Time to Onset of Meaningful Pain Relief
Description: Participants evaluated time to meaningful relief by stopping a second stopwatch labelled as "meaningful relief" at the moment they first began to experience meaningful relief. Stopwatch was active up to 12 hours after dosing or until stopped by participant, or participant became treatment failure prior to depressing the second stopwatch. Treatment failure was defined as participant taking rescue medication, or discontinuing due to lack of efficacy.
Time Frame: 0 to 12 hours post-dose
Population: FAS included all randomized participants who were dosed with the study medication and provided a baseline assessment. Here, "number of participants analyzed" signifies those participants who had the event (meaningful pain relief).
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Ibuprofen 250 mg + Acetaminophen 500 mg | Ibuprofen 250 mg | Acetaminophen 650 mg
Number analyzed (Participants) | 16 | 147 | 139 | 118
minutes | NA (8.8) [NA to NA] — Data was not estimable as median time to onset of meaningful relief was greater than (>) 720 minutes for placebo group. | 47.9 (9.2) [41.6 to 57.4] | 65.9 (8.9) [57.2 to 81.6] | 56.6 (8.8) [50.5 to 84.6]
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; p-value was calculated by using Gehan-Wilcoxon test, stratified by gender and baseline categorical PSR terms; Test type: Superiority or Other; p < 0.001, Gehan-Wilcoxon test
Statistical Analysis 2: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; p-value was calculated by using Gehan-Wilcoxon test, stratified by gender and baseline categorical PSR terms; Test type: Superiority or Other; p = 0.003, Gehan-Wilcoxon test
Statistical Analysis 3: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; p-value was calculated by using Gehan-Wilcoxon test, stratified by gender and baseline categorical PSR terms; Test type: Superiority or Other; p = 0.031, Gehan-Wilcoxon test
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen 250 mg; p-value was calculated by using Gehan-Wilcoxon test, stratified by gender and baseline categorical PSR terms; Test type: Superiority or Other; p < 0.001, Gehan-Wilcoxon test
Statistical Analysis 5: Comparison: Placebo vs Acetaminophen 650 mg; p-value was calculated by using Gehan-Wilcoxon test, stratified by gender and baseline categorical PSR terms; Test type: Superiority or Other; p < 0.001, Gehan-Wilcoxon test
Statistical Analysis 6: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; p-value was calculated by using Gehan-Wilcoxon test, stratified by gender and baseline categorical PSR terms; Test type: Superiority or Other; p = 0.631, Gehan-Wilcoxon test

7. Other Pre Specified Outcome: Time to Confirmed Onset of First Perceptible Relief
Description: Participants evaluated the time to first perceptible relief (confirmed by meaningful relief) by stopping the first stopwatch labeled 'first perceptible relief' at the moment they first began to experience any pain relief, if the participant also achieved meaningful relief by the end of the study. Stopwatch was active up to 12 hours after dosing or until stopped by the participant, or until the participant dropped out due to treatment failure prior to depressing the first stopwatch or until the time of withdrawal (discontinuation). Treatment failure was defined as participant taking rescue medication, or discontinuing due to lack of efficacy.
Time Frame: 0 to 12 hours post-dose
Population: FAS included all randomized participants who were dosed with the study medication and provided a baseline assessment. Here, "number of participants analyzed" signifies those participants who had the event (first perceptiblre relief).
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Ibuprofen 250 mg + Acetaminophen 500 mg | Ibuprofen 250 mg | Acetaminophen 650 mg
Number analyzed (Participants) | 16 | 149 | 139 | 118
minutes | NA (8.8) [NA to NA] — Data was not estimable as median time to confirmed onset of first perceptible relief was >720 minutes for placebo group. | 21.3 (9.2) [18.7 to 24.2] | 24.6 (8.9) [22.3 to 27.8] | 24.2 (8.8) [20.7 to 29.9]
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; p-value was calculated by using Gehan-Wilcoxon test, stratified by gender and baseline categorical PSR terms; Test type: Superiority or Other; p < 0.001, Gehan-Wilcoxon test
Statistical Analysis 2: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; p-value was calculated by using Gehan-Wilcoxon test, stratified by gender and baseline categorical PSR terms; Test type: Superiority or Other; p = 0.088, Gehan-Wilcoxon test
Statistical Analysis 3: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; p-value was calculated by using Gehan-Wilcoxon test, stratified by gender and baseline categorical PSR terms; Test type: Superiority or Other; p = 0.133, Gehan-Wilcoxon test
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen 250 mg; p-value was calculated by using Gehan-Wilcoxon test, stratified by gender and baseline categorical PSR terms; Test type: Superiority or Other; p < 0.001, Gehan-Wilcoxon test
Statistical Analysis 5: Comparison: Placebo vs Acetaminophen 650 mg; p-value was calculated by using Gehan-Wilcoxon test, stratified by gender and baseline categorical PSR terms; Test type: Superiority or Other; p < 0.001, Gehan-Wilcoxon test
Statistical Analysis 6: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; p-value was calculated by using Gehan-Wilcoxon test, stratified by gender and baseline categorical PSR terms; Test type: Superiority or Other; p = 0.887, Gehan-Wilcoxon test

8. Other Pre Specified Outcome: Pain Relief Rating (PRR) Score
Description: Participants answered a question: "how much relief do you have from your starting pain?" on a 5-point categorical pain relief rating scale. Scale ranges from 0= no relief to 4= complete relief.
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 hours post-dose
Population: FAS included all randomized participants who were dosed with the study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen 250 mg + Acetaminophen 500 mg | Ibuprofen 250 mg | Acetaminophen 650 mg
Number analyzed (Participants) | 56 | 172 | 175 | 165
units on a scale
  0.25 hour | 0.18 (0.39) | 0.51 (0.65) | 0.36 (0.61) | 0.50 (0.70)
  0.5 hour | 0.30 (0.46) | 1.29 (1.02) | 1.11 (0.97) | 1.20 (1.00)
  1 hour | 0.44 (0.63) | 2.19 (1.22) | 1.85 (1.18) | 1.86 (1.14)
  1.5 hour | 0.48 (0.74) | 2.47 (1.17) | 2.08 (1.25) | 1.90 (1.19)
  2 hour | 0.55 (0.96) | 2.65 (1.21) | 2.28 (1.33) | 1.86 (1.25)
  3 hour | 0.70 (1.09) | 2.75 (1.17) | 2.35 (1.36) | 1.66 (1.36)
  4 hour | 0.71 (1.16) | 2.71 (1.23) | 2.27 (1.39) | 1.55 (1.39)
  5 hour | 0.73 (1.21) | 2.64 (1.27) | 2.18 (1.37) | 1.50 (1.43)
  6 hour | 0.80 (1.31) | 2.36 (1.37) | 2.01 (1.42) | 1.29 (1.43)
  7 hour | 0.77 (1.31) | 2.04 (1.45) | 1.68 (1.43) | 1.14 (1.39)
  8 hour | 0.73 (1.24) | 1.75 (1.47) | 1.40 (1.41) | 1.03 (1.37)
  9 hour | 0.73 (1.23) | 1.41 (1.49) | 1.31 (1.45) | 0.95 (1.31)
  10 hour | 0.75 (1.24) | 1.20 (1.47) | 1.19 (1.43) | 0.95 (1.37)
  11 hour | 0.78 (1.29) | 1.06 (1.43) | 1.03 (1.40) | 0.88 (1.34)
  12 hour | 0.75 (1.25) | 0.97 (1.35) | 0.97 (1.40) | 0.85 (1.35)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 0.25 hour: Treatment difference and 95% CI were based on LS Mean from ANOVA with treatment, gender and baseline categorical PSR; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.33, 95% CI 2-sided [0.14 to 0.52]
Statistical Analysis 2: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.034, ANOVA; LS Mean Difference = 0.15, 95% CI 2-sided [0.01 to 0.28]
Statistical Analysis 3: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.963, ANOVA; LS Mean Difference = 0.00, 95% CI 2-sided [-0.13 to 0.14]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.062, ANOVA; LS Mean Difference = 0.18, 95% CI 2-sided [-0.01 to 0.37]
Statistical Analysis 5: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.001, ANOVA; LS Mean Difference = 0.32, 95% CI 2-sided [0.13 to 0.52]
Statistical Analysis 6: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.040, ANOVA; LS Mean Difference = -0.14, 95% CI 2-sided [-0.28 to -0.01]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 0.5 hour: Treatment difference and 95% CI were based on LS Mean from ANOVA with treatment, gender and baseline categorical PSR; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.99, 95% CI 2-sided [0.70 to 1.27]
Statistical Analysis 8: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 7]; Test type: Superiority or Other; p = 0.095, ANOVA; LS Mean Difference = 0.17, 95% CI 2-sided [-0.03 to 0.37]
Statistical Analysis 9: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 7]; Test type: Superiority or Other; p = 0.414, ANOVA; LS Mean Difference = 0.09, 95% CI 2-sided [-0.12 to 0.29]
Statistical Analysis 10: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 7]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.81, 95% CI 2-sided [0.52 to 1.10]
Statistical Analysis 11: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 7]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.90, 95% CI 2-sided [0.61 to 1.19]
Statistical Analysis 12: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 7]; Test type: Superiority or Other; p = 0.406, ANOVA; LS Mean Difference = -0.09, 95% CI 2-sided [-0.29 to 0.12]
Statistical Analysis 13: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 1 hour: Treatment difference and 95% CI were based on LS Mean from ANOVA with treatment, gender and baseline categorical PSR; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.75, 95% CI 2-sided [1.40 to 2.09]
Statistical Analysis 14: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 13]; Test type: Superiority or Other; p = 0.006, ANOVA; LS Mean Difference = 0.34, 95% CI 2-sided [0.10 to 0.58]
Statistical Analysis 15: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 13]; Test type: Superiority or Other; p = 0.009, ANOVA; LS Mean Difference = 0.33, 95% CI 2-sided [0.08 to 0.57]
Statistical Analysis 16: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 13]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.41, 95% CI 2-sided [1.07 to 1.75]
Statistical Analysis 17: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 13]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.42, 95% CI 2-sided [1.08 to 1.77]
Statistical Analysis 18: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 13]; Test type: Superiority or Other; p = 0.908, ANOVA; LS Mean Difference = -0.01, 95% CI 2-sided [-0.26 to 0.23]
Statistical Analysis 19: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 1.5 hour: Treatment difference and 95% CI were based on LS Mean from ANOVA with treatment, gender and baseline categorical PSR; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.99, 95% CI 2-sided [1.64 to 2.35]
Statistical Analysis 20: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 19]; Test type: Superiority or Other; p = 0.002, ANOVA; LS Mean Difference = 0.39, 95% CI 2-sided [0.15 to 0.64]
Statistical Analysis 21: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 19]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.57, 95% CI 2-sided [0.32 to 0.82]
Statistical Analysis 22: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 19]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.60, 95% CI 2-sided [1.25 to 1.95]
Statistical Analysis 23: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 19]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.42, 95% CI 2-sided [1.07 to 1.78]
Statistical Analysis 24: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 19]; Test type: Superiority or Other; p = 0.157, ANOVA; LS Mean Difference = 0.18, 95% CI 2-sided [-0.07 to 0.43]
Statistical Analysis 25: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 2 hour: Treatment difference and 95% CI were based on LS Mean from ANOVA with treatment, gender and baseline categorical PSR; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 2.10, 95% CI 2-sided [1.73 to 2.48]
Statistical Analysis 26: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 25]; Test type: Superiority or Other; p = 0.005, ANOVA; LS Mean Difference = 0.37, 95% CI 2-sided [0.11 to 0.63]
Statistical Analysis 27: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 25]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.79, 95% CI 2-sided [0.52 to 1.05]
Statistical Analysis 28: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 25]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.73, 95% CI 2-sided [1.36 to 2.10]
Statistical Analysis 29: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 25]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.31, 95% CI 2-sided [0.94 to 1.69]
Statistical Analysis 30: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 25]; Test type: Superiority or Other; p = 0.002, ANOVA; LS Mean Difference = 0.42, 95% CI 2-sided [0.15 to 0.68]
Statistical Analysis 31: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 3 hour: Treatment difference and 95% CI were based on LS Mean from ANOVA with treatment, gender and baseline categorical PSR; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 2.06, 95% CI 2-sided [1.67 to 2.45]
Statistical Analysis 32: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 31]; Test type: Superiority or Other; p = 0.004, ANOVA; LS Mean Difference = 0.40, 95% CI 2-sided [0.13 to 0.67]
Statistical Analysis 33: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 31]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.09, 95% CI 2-sided [0.82 to 1.37]
Statistical Analysis 34: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 31]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.66, 95% CI 2-sided [1.27 to 2.04]
Statistical Analysis 35: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 31]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.97, 95% CI 2-sided [0.58 to 1.36]
Statistical Analysis 36: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 31]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.69, 95% CI 2-sided [0.42 to 0.96]
Statistical Analysis 37: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 4 hour: Treatment difference and 95% CI were based on LS Mean from ANOVA with treatment, gender and baseline categorical PSR; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 2.00, 95% CI 2-sided [1.60 to 2.40]
Statistical Analysis 38: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 37]; Test type: Superiority or Other; p = 0.002, ANOVA; LS Mean Difference = 0.44, 95% CI 2-sided [0.16 to 0.72]
Statistical Analysis 39: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 37]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.16, 95% CI 2-sided [0.88 to 1.44]
Statistical Analysis 40: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 37]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.56, 95% CI 2-sided [1.16 to 1.96]
Statistical Analysis 41: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 37]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.84, 95% CI 2-sided [0.44 to 1.24]
Statistical Analysis 42: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 37]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.72, 95% CI 2-sided [0.44 to 1.00]
Statistical Analysis 43: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 5 hour: Treatment difference and 95% CI were based on LS Mean from ANOVA with treatment, gender and baseline categorical PSR; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.91, 95% CI 2-sided [1.50 to 2.31]
Statistical Analysis 44: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 43]; Test type: Superiority or Other; p = 0.001, ANOVA; LS Mean Difference = 0.46, 95% CI 2-sided [0.18 to 0.74]
Statistical Analysis 45: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 43]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.14, 95% CI 2-sided [0.85 to 1.43]
Statistical Analysis 46: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 43]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.45, 95% CI 2-sided [1.04 to 1.85]
Statistical Analysis 47: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 43]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.77, 95% CI 2-sided [0.36 to 1.17]
Statistical Analysis 48: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 43]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.68, 95% CI 2-sided [0.39 to 0.97]
Statistical Analysis 49: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 6 hour: Treatment difference and 95% CI were based on LS Mean from ANOVA with treatment, gender and baseline categorical PSR; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.55, 95% CI 2-sided [1.13 to 1.98]
Statistical Analysis 50: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 49]; Test type: Superiority or Other; p = 0.017, ANOVA; LS Mean Difference = 0.36, 95% CI 2-sided [0.06 to 0.65]
Statistical Analysis 51: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 49]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.07, 95% CI 2-sided [0.77 to 1.37]
Statistical Analysis 52: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 49]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.20, 95% CI 2-sided [0.78 to 1.62]
Statistical Analysis 53: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 49]; Test type: Superiority or Other; p = 0.026, ANOVA; LS Mean Difference = 0.48, 95% CI 2-sided [0.06 to 0.91]
Statistical Analysis 54: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 49]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.72, 95% CI 2-sided [0.42 to 1.01]
Statistical Analysis 55: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 7 hour: Treatment difference and 95% CI were based on LS Mean from ANOVA with treatment, gender and baseline categorical PSR; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.27, 95% CI 2-sided [0.84 to 1.69]
Statistical Analysis 56: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 55]; Test type: Superiority or Other; p = 0.017, ANOVA; LS Mean Difference = 0.36, 95% CI 2-sided [0.07 to 0.66]
Statistical Analysis 57: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 55]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.90, 95% CI 2-sided [0.60 to 1.20]
Statistical Analysis 58: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 55]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.90, 95% CI 2-sided [0.48 to 1.33]
Statistical Analysis 59: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 55]; Test type: Superiority or Other; p = 0.089, ANOVA; LS Mean Difference = 0.37, 95% CI 2-sided [-0.06 to 0.80]
Statistical Analysis 60: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 55]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.53, 95% CI 2-sided [0.24 to 0.83]
Statistical Analysis 61: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 8 hour: Treatment difference and 95% CI were based on LS Mean from ANOVA with treatment, gender and baseline categorical PSR; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.02, 95% CI 2-sided [0.60 to 1.44]
Statistical Analysis 62: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 61]; Test type: Superiority or Other; p = 0.018, ANOVA; LS Mean Difference = 0.35, 95% CI 2-sided [0.06 to 0.65]
Statistical Analysis 63: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 61]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.72, 95% CI 2-sided [0.42 to 1.02]
Statistical Analysis 64: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 61]; Test type: Superiority or Other; p = 0.002, ANOVA; LS Mean Difference = 0.67, 95% CI 2-sided [0.25 to 1.09]
Statistical Analysis 65: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 61]; Test type: Superiority or Other; p = 0.163, ANOVA; LS Mean Difference = 0.30, 95% CI 2-sided [-0.12 to 0.72]
Statistical Analysis 66: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 61]; Test type: Superiority or Other; p = 0.016, ANOVA; LS Mean Difference = 0.37, 95% CI 2-sided [0.07 to 0.66]
Statistical Analysis 67: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 9 hour: Treatment difference and 95% CI were based on LS Mean from ANOVA with treatment, gender and baseline categorical PSR; Test type: Superiority or Other; p = 0.002, ANOVA; LS Mean Difference = 0.68, 95% CI 2-sided [0.26 to 1.10]
Statistical Analysis 68: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 67]; Test type: Superiority or Other; p = 0.496, ANOVA; LS Mean Difference = 0.10, 95% CI 2-sided [-0.19 to 0.40]
Statistical Analysis 69: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 67]; Test type: Superiority or Other; p = 0.003, ANOVA; LS Mean Difference = 0.46, 95% CI 2-sided [0.16 to 0.76]
Statistical Analysis 70: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 67]; Test type: Superiority or Other; p = 0.008, ANOVA; LS Mean Difference = 0.57, 95% CI 2-sided [0.15 to 1.00]
Statistical Analysis 71: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 67]; Test type: Superiority or Other; p = 0.315, ANOVA; LS Mean Difference = 0.22, 95% CI 2-sided [-0.21 to 0.64]
Statistical Analysis 72: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 67]; Test type: Superiority or Other; p = 0.019, ANOVA; LS Mean Difference = 0.36, 95% CI 2-sided [0.06 to 0.66]
Statistical Analysis 73: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 10 hour: Treatment difference and 95% CI were based on LS Mean from ANOVA with treatment, gender and baseline categorical PSR; Test type: Superiority or Other; p = 0.038, ANOVA; LS Mean Difference = 0.45, 95% CI 2-sided [0.02 to 0.87]
Statistical Analysis 74: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 73]; Test type: Superiority or Other; p = 0.918, ANOVA; LS Mean Difference = 0.02, 95% CI 2-sided [-0.28 to 0.31]
Statistical Analysis 75: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 73]; Test type: Superiority or Other; p = 0.105, ANOVA; LS Mean Difference = 0.25, 95% CI 2-sided [-0.05 to 0.55]
Statistical Analysis 76: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 73]; Test type: Superiority or Other; p = 0.045, ANOVA; LS Mean Difference = 0.43, 95% CI 2-sided [0.01 to 0.85]
Statistical Analysis 77: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 73]; Test type: Superiority or Other; p = 0.355, ANOVA; LS Mean Difference = 0.20, 95% CI 2-sided [-0.22 to 0.62]
Statistical Analysis 78: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 73]; Test type: Superiority or Other; p = 0.127, ANOVA; LS Mean Difference = 0.23, 95% CI 2-sided [-0.07 to 0.53]
Statistical Analysis 79: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 11 hour: Treatment difference and 95% CI were based on LS Mean from ANOVA with treatment, gender and baseline categorical PSR; Test type: Superiority or Other; p = 0.171, ANOVA; LS Mean Difference = 0.29, 95% CI 2-sided [-0.12 to 0.70]
Statistical Analysis 80: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 79]; Test type: Superiority or Other; p = 0.790, ANOVA; LS Mean Difference = 0.04, 95% CI 2-sided [-0.25 to 0.33]
Statistical Analysis 81: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 79]; Test type: Superiority or Other; p = 0.235, ANOVA; LS Mean Difference = 0.18, 95% CI 2-sided [-0.12 to 0.47]
Statistical Analysis 82: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 79]; Test type: Superiority or Other; p = 0.236, ANOVA; LS Mean Difference = 0.25, 95% CI 2-sided [-0.16 to 0.66]
Statistical Analysis 83: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 79]; Test type: Superiority or Other; p = 0.599, ANOVA; LS Mean Difference = 0.11, 95% CI 2-sided [-0.30 to 0.53]
Statistical Analysis 84: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 79]; Test type: Superiority or Other; p = 0.353, ANOVA; LS Mean Difference = 0.14, 95% CI 2-sided [-0.15 to 0.43]
Statistical Analysis 85: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 12 hour: Treatment difference and 95% CI were based on LS Mean from ANOVA with treatment, gender and baseline categorical PSR; Test type: Superiority or Other; p = 0.293, ANOVA; LS Mean Difference = 0.22, 95% CI 2-sided [-0.19 to 0.62]
Statistical Analysis 86: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 85]; Test type: Superiority or Other; p = 0.986, ANOVA; LS Mean Difference = -0.00, 95% CI 2-sided [-0.28 to 0.28]
Statistical Analysis 87: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 85]; Test type: Superiority or Other; p = 0.459, ANOVA; LS Mean Difference = 0.11, 95% CI 2-sided [-0.18 to 0.39]
Statistical Analysis 88: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 85]; Test type: Superiority or Other; p = 0.287, ANOVA; LS Mean Difference = 0.22, 95% CI 2-sided [-0.18 to 0.62]
Statistical Analysis 89: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 85]; Test type: Superiority or Other; p = 0.600, ANOVA; LS Mean Difference = 0.11, 95% CI 2-sided [-0.30 to 0.51]
Statistical Analysis 90: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 85]; Test type: Superiority or Other; p = 0.447, ANOVA; LS Mean Difference = 0.11, 95% CI 2-sided [-0.17 to 0.40]

9. Other Pre Specified Outcome: Pain Intensity Difference on 11-Point Numerical Scale (PID11)
Description: PID11: baseline pain severity score minus pain severity score at a given time point. Pain intensity was assessed on an 11-point numerical pain severity rating scale. PID11 was calculated by subtracting the pain intensity score at given post-dose time points (pain severity score range: 0 =no pain to 10 =worst possible pain) from the baseline pain intensity scores (score range: 5 =moderate pain to 10 =worst possible pain; as participants with baseline pain score of at least moderate were included in study). Total possible score range for PID11: -5 (worst score) to 10 (best score).
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 hours post-dose
Population: FAS included all randomized participants who were dosed with the study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen 250 mg + Acetaminophen 500 mg | Ibuprofen 250 mg | Acetaminophen 650 mg
Number analyzed (Participants) | 56 | 172 | 175 | 165
units on a scale
  0.25 hour | 0.0 (0.9) | 0.6 (1.2) | 0.5 (1.2) | 0.7 (1.3)
  0.5 hour | 0.2 (1.2) | 2.2 (2.2) | 1.8 (2.0) | 2.0 (2.0)
  1 hour | 0.2 (1.6) | 4.1 (2.6) | 3.3 (2.6) | 3.3 (2.4)
  1.5 hour | 0.1 (1.8) | 4.8 (2.7) | 3.9 (2.8) | 3.4 (2.6)
  2 hour | 0.2 (2.1) | 5.1 (2.7) | 4.3 (3.0) | 3.3 (2.7)
  3 hour | 0.6 (2.6) | 5.3 (2.7) | 4.5 (3.1) | 2.9 (2.9)
  4 hour | 0.6 (2.7) | 5.2 (2.8) | 4.3 (3.0) | 2.7 (3.1)
  5 hour | 0.7 (2.9) | 5.0 (2.9) | 4.2 (3.1) | 2.6 (3.1)
  6 hour | 0.7 (3.0) | 4.4 (3.0) | 3.8 (3.1) | 2.2 (3.1)
  7 hour | 0.6 (3.0) | 3.8 (3.3) | 3.1 (3.1) | 1.8 (3.0)
  8 hour | 0.6 (2.9) | 3.1 (3.3) | 2.6 (3.0) | 1.6 (3.0)
  9 hour | 0.6 (2.8) | 2.4 (3.2) | 2.3 (3.0) | 1.4 (2.9)
  10 hour | 0.7 (2.9) | 2.0 (3.1) | 1.9 (2.9) | 1.4 (3.0)
  11 hour | 0.7 (2.9) | 1.7 (3.0) | 1.6 (2.9) | 1.3 (2.9)
  12 hour | 0.7 (2.9) | 1.5 (2.9) | 1.6 (2.9) | 1.2 (2.8)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 0.25 hour: Treatment difference and 95% CI were based on LS Mean from ANCOVA with treatment, gender, baseline categorical PSR as classification variables and baseline numerical PSR used as a continuous covariate; Test type: Superiority or Other; p = 0.001, ANCOVA; LS Mean Difference = 0.59, 95% CI 2-sided [0.23 to 0.96]
Statistical Analysis 2: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.297, ANCOVA; LS Mean Difference = 0.13, 95% CI 2-sided [-0.12 to 0.39]
Statistical Analysis 3: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.457, ANCOVA; LS Mean Difference = -0.10, 95% CI 2-sided [-0.35 to 0.16]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.012, ANCOVA; LS Mean Difference = 0.46, 95% CI 2-sided [0.10 to 0.82]
Statistical Analysis 5: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 0.69, 95% CI 2-sided [0.33 to 1.06]
Statistical Analysis 6: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.076, ANCOVA; LS Mean Difference = -0.23, 95% CI 2-sided [-0.49 to 0.02]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 0.5 hour: Treatment difference and 95% CI were based on LS Mean from ANCOVA with treatment, gender, baseline categorical PSR as classification variables and baseline numerical PSR used as a continuous covariate; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 2.03, 95% CI 2-sided [1.42 to 2.63]
Statistical Analysis 8: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 9, analysis 7]; Test type: Superiority or Other; p = 0.016, ANCOVA; LS Mean Difference = 0.51, 95% CI 2-sided [0.10 to 0.93]
Statistical Analysis 9: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 7]; Test type: Superiority or Other; p = 0.330, ANCOVA; LS Mean Difference = 0.21, 95% CI 2-sided [-0.21 to 0.64]
Statistical Analysis 10: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 9, analysis 7]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 1.51, 95% CI 2-sided [0.91 to 2.11]
Statistical Analysis 11: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 7]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 1.81, 95% CI 2-sided [1.21 to 2.42]
Statistical Analysis 12: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 7]; Test type: Superiority or Other; p = 0.163, ANCOVA; LS Mean Difference = -0.30, 95% CI 2-sided [-0.73 to 0.12]
Statistical Analysis 13: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 1 hour: Treatment difference and 95% CI were based on LS Mean from ANCOVA with treatment, gender, baseline categorical PSR as classification variables and baseline numerical PSR used as a continuous covariate; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 3.91, 95% CI 2-sided [3.18 to 4.65]
Statistical Analysis 14: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 9, analysis 13]; Test type: Superiority or Other; p = 0.001, ANCOVA; LS Mean Difference = 0.86, 95% CI 2-sided [0.35 to 1.38]
Statistical Analysis 15: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 13]; Test type: Superiority or Other; p = 0.003, ANCOVA; LS Mean Difference = 0.78, 95% CI 2-sided [0.26 to 1.31]
Statistical Analysis 16: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 9, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 3.05, 95% CI 2-sided [2.32 to 3.79]
Statistical Analysis 17: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 3.13, 95% CI 2-sided [2.39 to 3.87]
Statistical Analysis 18: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 13]; Test type: Superiority or Other; p = 0.769, ANCOVA; LS Mean Difference = -0.08, 95% CI 2-sided [-0.60 to 0.44]
Statistical Analysis 19: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 1.5 hour: Treatment difference and 95% CI were based on LS Mean from ANCOVA with treatment, gender, baseline categorical PSR as classification variables and baseline numerical PSR used as a continuous covariate; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 4.65, 95% CI 2-sided [3.88 to 5.42]
Statistical Analysis 20: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 9, analysis 19]; Test type: Superiority or Other; p = 0.002, ANCOVA; LS Mean Difference = 0.86, 95% CI 2-sided [0.32 to 1.40]
Statistical Analysis 21: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 19]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 1.38, 95% CI 2-sided [0.83 to 1.93]
Statistical Analysis 22: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 9, analysis 19]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 3.79, 95% CI 2-sided [3.02 to 4.56]
Statistical Analysis 23: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 19]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 3.27, 95% CI 2-sided [2.49 to 4.04]
Statistical Analysis 24: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 19]; Test type: Superiority or Other; p = 0.062, ANCOVA; LS Mean Difference = 0.52, 95% CI 2-sided [-0.03 to 1.06]
Statistical Analysis 25: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 2 hour: Treatment difference and 95% CI were based on LS Mean from ANCOVA with treatment, gender, baseline categorical PSR as classification variables and baseline numerical PSR used as a continuous covariate; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 4.83, 95% CI 2-sided [4.01 to 5.64]
Statistical Analysis 26: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 9, analysis 25]; Test type: Superiority or Other; p = 0.009, ANCOVA; LS Mean Difference = 0.76, 95% CI 2-sided [0.19 to 1.33]
Statistical Analysis 27: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 25]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 1.75, 95% CI 2-sided [1.17 to 2.33]
Statistical Analysis 28: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 9, analysis 25]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 4.06, 95% CI 2-sided [3.25 to 4.88]
Statistical Analysis 29: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 25]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 3.08, 95% CI 2-sided [2.26 to 3.90]
Statistical Analysis 30: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 25]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 0.98, 95% CI 2-sided [0.41 to 1.56]
Statistical Analysis 31: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 3 hour: Treatment difference and 95% CI were based on LS Mean from ANCOVA with treatment, gender, baseline categorical PSR as classification variables and baseline numerical PSR used as a continuous covariate; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 4.67, 95% CI 2-sided [3.82 to 5.52]
Statistical Analysis 32: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 9, analysis 31]; Test type: Superiority or Other; p = 0.010, ANCOVA; LS Mean Difference = 0.78, 95% CI 2-sided [0.19 to 1.38]
Statistical Analysis 33: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 31]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 2.41, 95% CI 2-sided [1.81 to 3.01]
Statistical Analysis 34: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 9, analysis 31]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 3.89, 95% CI 2-sided [3.04 to 4.74]
Statistical Analysis 35: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 31]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 2.26, 95% CI 2-sided [1.40 to 3.11]
Statistical Analysis 36: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 31]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 1.63, 95% CI 2-sided [1.02 to 2.23]
Statistical Analysis 37: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 4 hour: Treatment difference and 95% CI were based on LS Mean from ANCOVA with treatment, gender, baseline categorical PSR as classification variables and baseline numerical PSR used as a continuous covariate; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 4.53, 95% CI 2-sided [3.65 to 5.40]
Statistical Analysis 38: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 9, analysis 37]; Test type: Superiority or Other; p = 0.009, ANCOVA; LS Mean Difference = 0.82, 95% CI 2-sided [0.21 to 1.43]
Statistical Analysis 39: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 37]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 2.42, 95% CI 2-sided [1.79 to 3.04]
Statistical Analysis 40: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 9, analysis 37]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 3.71, 95% CI 2-sided [2.83 to 4.58]
Statistical Analysis 41: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 37]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 2.11, 95% CI 2-sided [1.23 to 2.99]
Statistical Analysis 42: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 37]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 1.60, 95% CI 2-sided [0.97 to 2.22]
Statistical Analysis 43: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 5 hour: Treatment difference and 95% CI were based on LS Mean from ANCOVA with treatment, gender, baseline categorical PSR as classification variables and baseline numerical PSR used as a continuous covariate; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 4.27, 95% CI 2-sided [3.37 to 5.17]
Statistical Analysis 44: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 9, analysis 43]; Test type: Superiority or Other; p = 0.012, ANCOVA; LS Mean Difference = 0.81, 95% CI 2-sided [0.18 to 1.44]
Statistical Analysis 45: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 43]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 2.36, 95% CI 2-sided [1.72 to 3.00]
Statistical Analysis 46: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 9, analysis 43]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 3.47, 95% CI 2-sided [2.57 to 4.36]
Statistical Analysis 47: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 43]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 1.91, 95% CI 2-sided [1.00 to 2.82]
Statistical Analysis 48: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 43]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 1.55, 95% CI 2-sided [0.92 to 2.19]
Statistical Analysis 49: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 6 hour: Treatment difference and 95% CI were based on LS Mean from ANCOVA with treatment, gender, baseline categorical PSR as classification variables and baseline numerical PSR used as a continuous covariate; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 3.68, 95% CI 2-sided [2.76 to 4.60]
Statistical Analysis 50: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 9, analysis 49]; Test type: Superiority or Other; p = 0.055, ANCOVA; LS Mean Difference = 0.63, 95% CI 2-sided [-0.01 to 1.27]
Statistical Analysis 51: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 49]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 2.19, 95% CI 2-sided [1.54 to 2.84]
Statistical Analysis 52: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 9, analysis 49]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 3.05, 95% CI 2-sided [2.14 to 3.97]
Statistical Analysis 53: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 49]; Test type: Superiority or Other; p = 0.002, ANCOVA; LS Mean Difference = 1.49, 95% CI 2-sided [0.57 to 2.42]
Statistical Analysis 54: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 49]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 1.56, 95% CI 2-sided [0.91 to 2.21]
Statistical Analysis 55: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 7 hour: Treatment difference and 95% CI were based on LS Mean from ANCOVA with treatment, gender, baseline categorical PSR as classification variables and baseline numerical PSR used as a continuous covariate; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 3.10, 95% CI 2-sided [2.17 to 4.03]
Statistical Analysis 56: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 9, analysis 55]; Test type: Superiority or Other; p = 0.049, ANCOVA; LS Mean Difference = 0.65, 95% CI 2-sided [0.00 to 1.30]
Statistical Analysis 57: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 55]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 1.93, 95% CI 2-sided [1.27 to 2.59]
Statistical Analysis 58: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 9, analysis 55]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 2.44, 95% CI 2-sided [1.52 to 3.37]
Statistical Analysis 59: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 55]; Test type: Superiority or Other; p = 0.015, ANCOVA; LS Mean Difference = 1.17, 95% CI 2-sided [0.23 to 2.10]
Statistical Analysis 60: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 55]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 1.28, 95% CI 2-sided [0.62 to 1.94]
Statistical Analysis 61: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 8 hour: Treatment difference and 95% CI were based on LS Mean from ANCOVA with treatment, gender, baseline categorical PSR as classification variables and baseline numerical PSR used as a continuous covariate; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 2.48, 95% CI 2-sided [1.56 to 3.40]
Statistical Analysis 62: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 9, analysis 61]; Test type: Superiority or Other; p = 0.087, ANCOVA; LS Mean Difference = 0.56, 95% CI 2-sided [-0.08 to 1.20]
Statistical Analysis 63: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 61]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 1.47, 95% CI 2-sided [0.82 to 2.12]
Statistical Analysis 64: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 9, analysis 61]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 1.92, 95% CI 2-sided [1.00 to 2.84]
Statistical Analysis 65: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 61]; Test type: Superiority or Other; p = 0.032, ANCOVA; LS Mean Difference = 1.01, 95% CI 2-sided [0.09 to 1.94]
Statistical Analysis 66: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 61]; Test type: Superiority or Other; p = 0.006, ANCOVA; LS Mean Difference = 0.91, 95% CI 2-sided [0.26 to 1.56]
Statistical Analysis 67: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 9 hour: Treatment difference and 95% CI were based on LS Mean from ANCOVA with treatment, gender, baseline categorical PSR as classification variables and baseline numerical PSR used as a continuous covariate; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 1.75, 95% CI 2-sided [0.85 to 2.66]
Statistical Analysis 68: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 9, analysis 67]; Test type: Superiority or Other; p = 0.669, ANCOVA; LS Mean Difference = 0.14, 95% CI 2-sided [-0.49 to 0.77]
Statistical Analysis 69: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 67]; Test type: Superiority or Other; p = 0.007, ANCOVA; LS Mean Difference = 0.89, 95% CI 2-sided [0.24 to 1.53]
Statistical Analysis 70: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 9, analysis 67]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 1.61, 95% CI 2-sided [0.71 to 2.52]
Statistical Analysis 71: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 67]; Test type: Superiority or Other; p = 0.063, ANCOVA; LS Mean Difference = 0.86, 95% CI 2-sided [-0.05 to 1.78]
Statistical Analysis 72: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 67]; Test type: Superiority or Other; p = 0.022, ANCOVA; LS Mean Difference = 0.75, 95% CI 2-sided [0.11 to 1.39]
Statistical Analysis 73: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 10 hour: Treatment difference and 95% CI were based on LS Mean from ANCOVA with treatment, gender, baseline categorical PSR as classification variables and baseline numerical PSR used as a continuous covariate; Test type: Superiority or Other; p = 0.008, ANCOVA; LS Mean Difference = 1.22, 95% CI 2-sided [0.32 to 2.12]
Statistical Analysis 74: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 9, analysis 73]; Test type: Superiority or Other; p = 0.876, ANCOVA; LS Mean Difference = 0.05, 95% CI 2-sided [-0.58 to 0.68]
Statistical Analysis 75: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 73]; Test type: Superiority or Other; p = 0.134, ANCOVA; LS Mean Difference = 0.49, 95% CI 2-sided [-0.15 to 1.13]
Statistical Analysis 76: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 9, analysis 73]; Test type: Superiority or Other; p = 0.011, ANCOVA; LS Mean Difference = 1.17, 95% CI 2-sided [0.27 to 2.07]
Statistical Analysis 77: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 73]; Test type: Superiority or Other; p = 0.112, ANCOVA; LS Mean Difference = 0.73, 95% CI 2-sided [-0.17 to 1.64]
Statistical Analysis 78: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 73]; Test type: Superiority or Other; p = 0.179, ANCOVA; LS Mean Difference = 0.44, 95% CI 2-sided [-0.20 to 1.08]
Statistical Analysis 79: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 11 hour: Treatment difference and 95% CI were based on LS Mean from ANCOVA with treatment, gender, baseline categorical PSR as classification variables and baseline numerical PSR used as a continuous covariate; Test type: Superiority or Other; p = 0.032, ANCOVA; LS Mean Difference = 0.97, 95% CI 2-sided [0.09 to 1.85]
Statistical Analysis 80: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 9, analysis 79]; Test type: Superiority or Other; p = 0.850, ANCOVA; LS Mean Difference = 0.06, 95% CI 2-sided [-0.56 to 0.67]
Statistical Analysis 81: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 79]; Test type: Superiority or Other; p = 0.311, ANCOVA; LS Mean Difference = 0.32, 95% CI 2-sided [-0.30 to 0.95]
Statistical Analysis 82: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 9, analysis 79]; Test type: Superiority or Other; p = 0.043, ANCOVA; LS Mean Difference = 0.91, 95% CI 2-sided [0.03 to 1.79]
Statistical Analysis 83: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 79]; Test type: Superiority or Other; p = 0.154, ANCOVA; LS Mean Difference = 0.64, 95% CI [-0.24 to 1.53]
Statistical Analysis 84: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 79]; Test type: Superiority or Other; p = 0.408, ANCOVA; LS Mean Difference = 0.26, 95% CI 2-sided [-0.36 to 0.89]
Statistical Analysis 85: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 12 hour: Treatment difference and 95% CI were based on LS Mean from ANCOVA with treatment, gender, baseline categorical PSR as classification variables and baseline numerical PSR used as a continuous covariate; Test type: Superiority or Other; p = 0.065, ANCOVA; LS Mean Difference = 0.81, 95% CI 2-sided [-0.05 to 1.68]
Statistical Analysis 86: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 9, analysis 85]; Test type: Superiority or Other; p = 0.862, ANCOVA; LS Mean Difference = -0.05, 95% CI 2-sided [-0.66 to 0.55]
Statistical Analysis 87: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 85]; Test type: Superiority or Other; p = 0.352, ANCOVA; LS Mean Difference = 0.29, 95% CI 2-sided [-0.32 to 0.90]
Statistical Analysis 88: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 9, analysis 85]; Test type: Superiority or Other; p = 0.049, ANCOVA; LS Mean Difference = 0.87, 95% CI 2-sided [0.00 to 1.73]
Statistical Analysis 89: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 85]; Test type: Superiority or Other; p = 0.239, ANCOVA; LS Mean Difference = 0.52, 95% CI 2-sided [-0.35 to 1.39]
Statistical Analysis 90: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 9, analysis 85]; Test type: Superiority or Other; p = 0.270, ANCOVA; LS Mean Difference = 0.34, 95% CI 2-sided [-0.27 to 0.96]

10. Other Pre Specified Outcome: Pain Intensity Difference on 4-Point Categorical Scale (PID4)
Description: PID4: baseline pain severity score minus pain severity score at a given time point. Pain intensity was assessed on a 4-point categorical pain severity rating scale. PID4 was calculated by subtracting the pain intensity score at given post-dose time points (pain severity score range: 0 [no pain] to 3 [worst possible pain]) from the baseline pain intensity scores (score range: 2 =moderate pain to 3 =worst possible pain; as participants with baseline pain score of at least moderate were included in study). Total possible score range for PID4: -1 (worst score) to 3 (best score).
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 hours post-dose
Population: FAS included all randomized participants who were dosed with the study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen 250 mg + Acetaminophen 500 mg | Ibuprofen 250 mg | Acetaminophen 650 mg
Number analyzed (Participants) | 56 | 172 | 175 | 165
units on a scale
  0.25 hour | 0.00 (0.27) | 0.15 (0.47) | 0.12 (0.47) | 0.20 (0.51)
  0.5 hour | 0.05 (0.40) | 0.60 (0.74) | 0.46 (0.72) | 0.61 (0.73)
  1 hour | 0.04 (0.54) | 1.18 (0.90) | 0.89 (0.95) | 0.98 (0.86)
  1.5 hour | 0.00 (0.57) | 1.36 (0.89) | 1.09 (1.01) | 0.98 (0.86)
  2 hour | 0.05 (0.75) | 1.47 (0.96) | 1.22 (1.09) | 0.92 (0.90)
  3 hour | 0.16 (0.83) | 1.55 (0.93) | 1.25 (1.09) | 0.81 (0.93)
  4 hour | 0.16 (0.87) | 1.15 (0.96) | 1.21 (1.08) | 0.74 (0.94)
  5 hour | 0.14 (0.88) | 1.44 (1.00) | 1.13 (1.05) | 0.75 (0.95)
  6 hour | 0.16 (0.93) | 1.27 (1.04) | 1.02 (1.04) | 0.63 (0.97)
  7 hour | 0.13 (0.88) | 1.04 (1.09) | 0.83 (1.02) | 0.50 (0.97)
  8 hour | 0.11 (0.82) | 0.88 (1.07) | 0.67 (0.97) | 0.45 (0.92)
  9 hour | 0.11 (0.82) | 0.69 (1.06) | 0.60 (0.95) | 0.36 (0.88)
  10 hour | 0.13 (0.85) | 0.52 (1.02) | 0.50 (0.95) | 0.37 (0.91)
  11 hour | 0.13 (0.85) | 0.45 (0.97) | 0.40 (0.93) | 0.32 (0.87)
  12 hour | 0.13 (0.85) | 0.38 (0.92) | 0.39 (0.96) | 0.27 (0.85)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.031, ANOVA; LS Mean Difference = 0.15, 95% CI 2-sided [0.01 to 0.28]
Statistical Analysis 2: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.527, ANOVA; LS Mean Difference = 0.03, 95% CI 2-sided [-0.06 to 0.12]
Statistical Analysis 3: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.386, ANOVA; LS Mean Difference = -0.04, 95% CI 2-sided [-0.14 to 0.05]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.084, ANOVA; LS Mean Difference = 0.12, 95% CI 2-sided [-0.02 to 0.25]
Statistical Analysis 5: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.006, ANOVA; LS Mean Difference = 0.19, 95% CI 2-sided [0.06 to 0.32]
Statistical Analysis 6: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.135, ANOVA; LS Mean Difference = -0.07, 95% CI 2-sided [-0.17 to 0.02]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 7]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.54, 95% CI 2-sided [0.34 to 0.73]
Statistical Analysis 8: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 7]; Test type: Superiority or Other; p = 0.062, ANOVA; LS Mean Difference = 0.13, 95% CI 2-sided [-0.01 to 0.27]
Statistical Analysis 9: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 7]; Test type: Superiority or Other; p = 0.977, ANOVA; LS Mean Difference = 0.00, 95% CI 2-sided [-0.14 to 0.14]
Statistical Analysis 10: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 7]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.41, 95% CI 2-sided [0.21 to 0.60]
Statistical Analysis 11: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 7]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.53, 95% CI 2-sided [0.34 to 0.73]
Statistical Analysis 12: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 7]; Test type: Superiority or Other; p = 0.069, ANOVA; LS Mean Difference = -0.13, 95% CI 2-sided [-0.27 to 0.01]
Statistical Analysis 13: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 13]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.14, 95% CI 2-sided [0.90 to 1.38]
Statistical Analysis 14: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 13]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.29, 95% CI 2-sided [0.12 to 0.46]
Statistical Analysis 15: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 13]; Test type: Superiority or Other; p = 0.011, ANOVA; LS Mean Difference = 0.22, 95% CI 2-sided [0.05 to 0.39]
Statistical Analysis 16: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 13]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.85, 95% CI 2-sided [0.61 to 1.09]
Statistical Analysis 17: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 13]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.92, 95% CI 2-sided [0.67 to 1.16]
Statistical Analysis 18: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 13]; Test type: Superiority or Other; p = 0.427, ANOVA; LS Mean Difference = -0.07, 95% CI 2-sided [-0.24 to 0.10]
Statistical Analysis 19: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 19]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.36, 95% CI 2-sided [1.11 to 1.60]
Statistical Analysis 20: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 19]; Test type: Superiority or Other; p = 0.002, ANOVA; LS Mean Difference = 0.27, 95% CI 2-sided [0.10 to 0.44]
Statistical Analysis 21: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 19]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.41, 95% CI 2-sided [0.23 to 0.58]
Statistical Analysis 22: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 19]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.09, 95% CI 2-sided [0.84 to 1.33]
Statistical Analysis 23: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 19]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.95, 95% CI 2-sided [0.70 to 1.20]
Statistical Analysis 24: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 19]; Test type: Superiority or Other; p = 0.123, ANOVA; LS Mean Difference = 0.14, 95% CI 2-sided [-0.04 to 0.31]
Statistical Analysis 25: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 25]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.40, 95% CI 2-sided [1.14 to 1.67]
Statistical Analysis 26: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 25]; Test type: Superiority or Other; p = 0.012, ANOVA; LS Mean Difference = 0.24, 95% CI 2-sided [0.05 to 0.42]
Statistical Analysis 27: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 25]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.56, 95% CI 2-sided [0.38 to 0.75]
Statistical Analysis 28: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 25]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.17, 95% CI 2-sided [0.90 to 1.43]
Statistical Analysis 29: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 25]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.84, 95% CI 2-sided [0.57 to 1.11]
Statistical Analysis 30: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 25]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.33, 95% CI 2-sided [0.14 to 0.51]
Statistical Analysis 31: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 31]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.38, 95% CI 2-sided [1.11 to 1.65]
Statistical Analysis 32: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 31]; Test type: Superiority or Other; p = 0.002, ANOVA; LS Mean Difference = 0.30, 95% CI 2-sided [0.11 to 0.48]
Statistical Analysis 33: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 31]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.76, 95% CI 2-sided [0.56 to 0.95]
Statistical Analysis 34: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 31]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.09, 95% CI 2-sided [0.82 to 1.36]
Statistical Analysis 35: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 31]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.63, 95% CI 2-sided [0.35 to 0.90]
Statistical Analysis 36: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 31]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.46, 95% CI 2-sided [0.27 to 0.65]
Statistical Analysis 37: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 37]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.34, 95% CI 2-sided [1.06 to 1.61]
Statistical Analysis 38: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 37]; Test type: Superiority or Other; p = 0.003, ANOVA; LS Mean Difference = 0.30, 95% CI 2-sided [0.10 to 0.49]
Statistical Analysis 39: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 37]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.78, 95% CI 2-sided [0.58 to 0.98]
Statistical Analysis 40: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 37]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.04, 95% CI 2-sided [0.76 to 1.32]
Statistical Analysis 41: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 37]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.56, 95% CI 2-sided [0.28 to 0.84]
Statistical Analysis 42: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 37]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.48, 95% CI 2-sided [0.29 to 0.68]
Statistical Analysis 43: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 43]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.28, 95% CI 2-sided [1.00 to 1.57]
Statistical Analysis 44: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 43]; Test type: Superiority or Other; p = 0.003, ANOVA; LS Mean Difference = 0.30, 95% CI 2-sided [0.10 to 0.50]
Statistical Analysis 45: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 43]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.71, 95% CI 2-sided [0.51 to 0.91]
Statistical Analysis 46: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 43]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.98, 95% CI 2-sided [0.70 to 1.27]
Statistical Analysis 47: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 43]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.58, 95% CI 2-sided [0.29 to 0.86]
Statistical Analysis 48: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 43]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.41, 95% CI 2-sided [0.21 to 0.61]
Statistical Analysis 49: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 49]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.10, 95% CI 2-sided [0.81 to 1.38]
Statistical Analysis 50: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 49]; Test type: Superiority or Other; p = 0.014, ANOVA; LS Mean Difference = 0.25, 95% CI 2-sided [0.05 to 0.45]
Statistical Analysis 51: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 49]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.66, 95% CI 2-sided [0.45 to 0.86]
Statistical Analysis 52: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 49]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.85, 95% CI 2-sided [0.56 to 1.13]
Statistical Analysis 53: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 49]; Test type: Superiority or Other; p = 0.003, ANOVA; LS Mean Difference = 0.44, 95% CI 2-sided [0.15 to 0.73]
Statistical Analysis 54: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 49]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.41, 95% CI 2-sided [0.21 to 0.61]
Statistical Analysis 55: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 55]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.91, 95% CI 2-sided [0.62 to 1.20]
Statistical Analysis 56: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 55]; Test type: Superiority or Other; p = 0.041, ANOVA; LS Mean Difference = 0.21, 95% CI 2-sided [0.01 to 0.42]
Statistical Analysis 57: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 55]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.56, 95% CI 2-sided [0.35 to 0.76]
Statistical Analysis 58: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 55]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.70, 95% CI 2-sided [0.41 to 0.99]
Statistical Analysis 59: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 55]; Test type: Superiority or Other; p = 0.018, ANOVA; LS Mean Difference = 0.35, 95% CI 2-sided [0.06 to 0.65]
Statistical Analysis 60: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 55]; Test type: Superiority or Other; p = 0.001, ANOVA; LS Mean Difference = 0.34, 95% CI 2-sided [0.14 to 0.55]
Statistical Analysis 61: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 61]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.76, 95% CI 2-sided [0.48 to 1.05]
Statistical Analysis 62: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 61]; Test type: Superiority or Other; p = 0.045, ANOVA; LS Mean Difference = 0.20, 95% CI 2-sided [0.00 to 0.40]
Statistical Analysis 63: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 61]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.44, 95% CI 2-sided [0.24 to 0.64]
Statistical Analysis 64: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 61]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.56, 95% CI 2-sided [0.28 to 0.84]
Statistical Analysis 65: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 61]; Test type: Superiority or Other; p = 0.027, ANOVA; LS Mean Difference = 0.32, 95% CI 2-sided [0.04 to 0.61]
Statistical Analysis 66: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 61]; Test type: Superiority or Other; p = 0.020, ANOVA; LS Mean Difference = 0.24, 95% CI 2-sided [0.04 to 0.44]
Statistical Analysis 67: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 67]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.57, 95% CI 2-sided [0.29 to 0.85]
Statistical Analysis 68: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 67]; Test type: Superiority or Other; p = 0.374, ANOVA; LS Mean Difference = 0.09, 95% CI 2-sided [-0.11 to 0.28]
Statistical Analysis 69: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 67]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.34, 95% CI 2-sided [0.14 to 0.54]
Statistical Analysis 70: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 67]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.48, 95% CI 2-sided [0.20 to 0.76]
Statistical Analysis 71: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 67]; Test type: Superiority or Other; p = 0.106, ANOVA; LS Mean Difference = 0.23, 95% CI 2-sided [-0.05 to 0.51]
Statistical Analysis 72: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 67]; Test type: Superiority or Other; p = 0.013, ANOVA; LS Mean Difference = 0.25, 95% CI 2-sided [0.05 to 0.45]
Statistical Analysis 73: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 73]; Test type: Superiority or Other; p = 0.006, ANOVA; LS Mean Difference = 0.39, 95% CI 2-sided [0.11 to 0.67]
Statistical Analysis 74: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 73]; Test type: Superiority or Other; p = 0.796, ANOVA; LS Mean Difference = 0.03, 95% CI 2-sided [-0.17 to 0.22]
Statistical Analysis 75: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 73]; Test type: Superiority or Other; p = 0.104, ANOVA; LS Mean Difference = 0.16, 95% CI 2-sided [-0.03 to 0.36]
Statistical Analysis 76: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 73]; Test type: Superiority or Other; p = 0.010, ANOVA; LS Mean Difference = 0.37, 95% CI 2-sided [0.09 to 0.65]
Statistical Analysis 77: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 73]; Test type: Superiority or Other; p = 0.114, ANOVA; LS Mean Difference = 0.23, 95% CI 2-sided [-0.05 to 0.51]
Statistical Analysis 78: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 73]; Test type: Superiority or Other; p = 0.168, ANOVA; LS Mean Difference = 0.14, 95% CI 2-sided [-0.06 to 0.34]
Statistical Analysis 79: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 79]; Test type: Superiority or Other; p = 0.022, ANOVA; LS Mean Difference = 0.32, 95% CI 2-sided [0.05 to 0.59]
Statistical Analysis 80: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 79]; Test type: Superiority or Other; p = 0.620, ANOVA; LS Mean Difference = 0.05, 95% CI 2-sided [-0.14 to 0.24]
Statistical Analysis 81: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 79]; Test type: Superiority or Other; p = 0.164, ANOVA; LS Mean Difference = 0.14, 95% CI 2-sided [-0.06 to 0.33]
Statistical Analysis 82: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 79]; Test type: Superiority or Other; p = 0.052, ANOVA; LS Mean Difference = 0.27, 95% CI 2-sided [-0.00 to 0.54]
Statistical Analysis 83: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 79]; Test type: Superiority or Other; p = 0.196, ANOVA; LS Mean Difference = 0.18, 95% CI 2-sided [-0.09 to 0.45]
Statistical Analysis 84: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 79]; Test type: Superiority or Other; p = 0.364, ANOVA; LS Mean Difference = 0.09, 95% CI 2-sided [-0.10 to 0.28]
Statistical Analysis 85: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 85]; Test type: Superiority or Other; p = 0.071, ANOVA; LS Mean Difference = 0.25, 95% CI 2-sided [-0.02 to 0.52]
Statistical Analysis 86: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 85]; Test type: Superiority or Other; p = 0.865, ANOVA; LS Mean Difference = -0.02, 95% CI [-0.20 to 0.17]
Statistical Analysis 87: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 85]; Test type: Superiority or Other; p = 0.238, ANOVA; LS Mean Difference = 0.11, 95% CI 2-sided [-0.08 to 0.30]
Statistical Analysis 88: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 85]; Test type: Superiority or Other; p = 0.054, ANOVA; LS Mean Difference = 0.26, 95% CI 2-sided [-0.00 to 0.53]
Statistical Analysis 89: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 85]; Test type: Superiority or Other; p = 0.335, ANOVA; LS Mean Difference = 0.13, 95% CI 2-sided [-0.14 to 0.40]
Statistical Analysis 90: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 85]; Test type: Superiority or Other; p = 0.176, ANOVA; LS Mean Difference = 0.13, 95% CI 2-sided [-0.06 to 0.32]

11. Other Pre Specified Outcome: Sum of Pain Relief Rating and Pain Intensity Difference on 4-Point Categorical Scale (PRID4)
Description: PRID4: sum of PID and PRR at each post-dose time points up to 12 hours. Score range for PRID: -1(worst score) to 7(best score). PID was calculated by subtracting the pain intensity score at given post-dose time points (pain severity score range: 0 [no pain] to 3 [worst possible pain]) from the baseline pain intensity scores (score range: 2 =moderate pain to 3 =worst possible pain; as participants with baseline pain score of at least moderate were included in study). Total possible score range for PID4: -1 (worst score) to 3 (best score). PRR was assessed on a 5-point categorical pain relief rating scale which ranges from 0 =no relief to 4 =complete relief.
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 hours post-dose
Population: FAS included all randomized participants who were dosed with the study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen 250 mg + Acetaminophen 500 mg | Ibuprofen 250 mg | Acetaminophen 650 mg
Number analyzed (Participants) | 56 | 172 | 175 | 165
units on a scale
  0.25 hour | 0.2 (0.5) | 0.7 (1.0) | 0.5 (1.0) | 0.7 (1.1)
  0.5 hour | 0.4 (0.7) | 1.9 (1.7) | 1.6 (1.6) | 1.8 (1.6)
  1 hour | 0.5 (1.0) | 3.4 (2.0) | 2.7 (2.0) | 2.8 (1.9)
  1.5 hour | 0.5 (1.2) | 3.8 (2.0) | 3.2 (2.2) | 2.9 (1.9)
  2 hour | 0.6 (1.6) | 4.1 (2.1) | 3.5 (2.4) | 2.8 (2.1)
  3 hour | 0.9 (1.8) | 4.3 (2.0) | 3.6 (2.4) | 2.5 (2.2)
  4 hour | 0.9 (1.9) | 4.2 (2.1) | 3.5 (2.4) | 2.3 (2.3)
  5 hour | 0.9 (2.0) | 4.1 (2.2) | 3.3 (2.4) | 2.2 (2.3)
  6 hour | 1.0 (2.2) | 3.6 (2.3) | 3.0 (2.4) | 1.9 (2.3)
  7 hour | 0.9 (2.1) | 3.1 (2.5) | 2.5 (2.4) | 1.6 (2.3)
  8 hour | 0.8 (2.0) | 2.6 (2.5) | 2.1 (2.3) | 1.5 (2.2)
  9 hour | 0.8 (2.0) | 2.1 (2.5) | 1.9 (2.3) | 1.3 (2.1)
  10 hour | 0.9 (2.0) | 1.7 (2.4) | 1.7 (2.3) | 1.3 (2.2)
  11 hour | 0.9 (2.1) | 1.5 (2.3) | 1.4 (2.3) | 1.2 (2.1)
  12 hour | 0.9 (2.0) | 1.3 (2.2) | 1.4 (2.3) | 1.1 (2.1)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.002, ANOVA; LS Mean Difference = 0.48, 95% CI 2-sided [0.18 to 0.77]
Statistical Analysis 2: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.098, ANOVA; LS Mean Difference = 0.18, 95% CI 2-sided [-0.03 to 0.38]
Statistical Analysis 3: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.719, ANOVA; LS Mean Difference = -0.04, 95% CI 2-sided [-0.25 to 0.17]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.048, ANOVA; LS Mean Difference = 0.30, 95% CI 2-sided [0.00 to 0.60]
Statistical Analysis 5: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.51, 95% CI 2-sided [0.21 to 0.81]
Statistical Analysis 6: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.046, ANOVA; LS Mean Difference = -0.21, 95% CI 2-sided [-0.42 to -0.00]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 7]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.52, 95% CI 2-sided [1.05 to 1.99]
Statistical Analysis 8: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 7]; Test type: Superiority or Other; p = 0.069, ANOVA; LS Mean Difference = 0.30, 95% CI 2-sided [-0.02 to 0.63]
Statistical Analysis 9: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 7]; Test type: Superiority or Other; p = 0.604, ANOVA; LS Mean Difference = 0.09, 95% CI 2-sided [-0.24 to 0.42]
Statistical Analysis 10: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 7]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.22, 95% CI 2-sided [0.75 to 1.69]
Statistical Analysis 11: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 7]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.43, 95% CI 2-sided [0.96 to 1.90]
Statistical Analysis 12: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 7]; Test type: Superiority or Other; p = 0.200, ANOVA; LS Mean Difference = -0.22, 95% CI 2-sided [-0.54 to 0.11]
Statistical Analysis 13: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 13]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 2.89, 95% CI 2-sided [2.32 to 3.46]
Statistical Analysis 14: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 13]; Test type: Superiority or Other; p = 0.002, ANOVA; LS Mean Difference = 0.63, 95% CI 2-sided [0.23 to 1.03]
Statistical Analysis 15: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 13]; Test type: Superiority or Other; p = 0.008, ANOVA; LS Mean Difference = 0.55, 95% CI 2-sided [0.14 to 0.95]
Statistical Analysis 16: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 13]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 2.26, 95% CI 2-sided [1.69 to 2.83]
Statistical Analysis 17: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 13]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 2.34, 95% CI 2-sided [1.77 to 2.91]
Statistical Analysis 18: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 13]; Test type: Superiority or Other; p = 0.685, ANOVA; LS Mean Difference = -0.08, 95% CI 2-sided [-0.49 to 0.32]
Statistical Analysis 19: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 19]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 3.35, 95% CI 2-sided [2.77 to 3.93]
Statistical Analysis 20: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 19]; Test type: Superiority or Other; p = 0.001, ANOVA; LS Mean Difference = 0.66, 95% CI 2-sided [0.26 to 1.07]
Statistical Analysis 21: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 19]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.98, 95% CI 2-sided [0.57 to 1.39]
Statistical Analysis 22: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 19]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 2.69, 95% CI 2-sided [2.11 to 3.27]
Statistical Analysis 23: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 19]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 2.37, 95% CI 2-sided [1.79 to 2.96]
Statistical Analysis 24: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 19]; Test type: Superiority or Other; p = 0.132, ANOVA; LS Mean Difference = 0.32, 95% CI 2-sided [-0.10 to 0.73]
Statistical Analysis 25: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 25]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 3.50, 95% CI 2-sided [2.88 to 4.13]
Statistical Analysis 26: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 25]; Test type: Superiority or Other; p = 0.007, ANOVA; LS Mean Difference = 0.61, 95% CI 2-sided [0.17 to 1.05]
Statistical Analysis 27: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 25]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.35, 95% CI 2-sided [0.91 to 1.80]
Statistical Analysis 28: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 25]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 2.90, 95% CI 2-sided [2.27 to 3.52]
Statistical Analysis 29: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 25]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 2.15, 95% CI 2-sided [1.52 to 2.79]
Statistical Analysis 30: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 25]; Test type: Superiority or Other; p = 0.001, ANOVA; LS Mean Difference = 0.74, 95% CI 2-sided [0.30 to 1.19]
Statistical Analysis 31: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 31]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 3.44, 95% CI 2-sided [2.79 to 4.09]
Statistical Analysis 32: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 31]; Test type: Superiority or Other; p = 0.003, ANOVA; LS Mean Difference = 0.70, 95% CI 2-sided [0.24 to 1.15]
Statistical Analysis 33: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 31]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.85, 95% CI 2-sided [1.39 to 2.31]
Statistical Analysis 34: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 31]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 2.74, 95% CI 2-sided [2.10 to 3.39]
Statistical Analysis 35: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 31]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.59, 95% CI 2-sided [0.94 to 2.24]
Statistical Analysis 36: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 31]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.15, 95% CI 2-sided [0.69 to 1.61]
Statistical Analysis 37: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 37]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 3.33, 95% CI 2-sided [2.67 to 4.00]
Statistical Analysis 38: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 37]; Test type: Superiority or Other; p = 0.002, ANOVA; LS Mean Difference = 0.74, 95% CI 2-sided [0.27 to 1.20]
Statistical Analysis 39: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 37]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.94, 95% CI 2-sided [1.47 to 2.41]
Statistical Analysis 40: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 37]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 2.60, 95% CI 2-sided [1.93 to 3.26]
Statistical Analysis 41: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 37]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.40, 95% CI 2-sided [0.73 to 2.07]
Statistical Analysis 42: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 37]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.20, 95% CI 2-sided [0.73 to 1.67]
Statistical Analysis 43: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 43]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 3.19, 95% CI 2-sided [2.51 to 3.87]
Statistical Analysis 44: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 43]; Test type: Superiority or Other; p = 0.002, ANOVA; LS Mean Difference = 0.76, 95% CI 2-sided [0.29 to 1.23]
Statistical Analysis 45: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 43]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.85, 95% CI 2-sided [1.37 to 2.33]
Statistical Analysis 46: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 43]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 2.43, 95% CI 2-sided [1.75 to 3.11]
Statistical Analysis 47: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 43]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.34, 95% CI 2-sided [0.66 to 2.03]
Statistical Analysis 48: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 43]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.09, 95% CI 2-sided [0.61 to 1.56]
Statistical Analysis 49: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 49]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 2.65, 95% CI 2-sided [1.95 to 3.35]
Statistical Analysis 50: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 49]; Test type: Superiority or Other; p = 0.015, ANOVA; LS Mean Difference = 0.61, 95% CI 2-sided [0.12 to 1.09]
Statistical Analysis 51: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 49]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.73, 95% CI 2-sided [1.24 to 2.22]
Statistical Analysis 52: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 49]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 2.05, 95% CI 2-sided [1.35 to 2.74]
Statistical Analysis 53: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 49]; Test type: Superiority or Other; p = 0.010, ANOVA; LS Mean Difference = 0.92, 95% CI 2-sided [0.22 to 1.62]
Statistical Analysis 54: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 49]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.12, 95% CI 2-sided [0.63 to 1.61]
Statistical Analysis 55: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 55]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 2.18, 95% CI 2-sided [1.47 to 2.88]
Statistical Analysis 56: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 55]; Test type: Superiority or Other; p = 0.022, ANOVA; LS Mean Difference = 0.57, 95% CI 2-sided [0.08 to 1.06]
Statistical Analysis 57: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 55]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.45, 95% CI 2-sided [0.95 to 1.95]
Statistical Analysis 58: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 55]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.60, 95% CI 2-sided [0.90 to 2.30]
Statistical Analysis 59: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 55]; Test type: Superiority or Other; p = 0.045, ANOVA; LS Mean Difference = 0.72, 95% CI 2-sided [0.02 to 1.43]
Statistical Analysis 60: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 55]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.88, 95% CI 2-sided [0.38 to 1.38]
Statistical Analysis 61: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 61]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.78, 95% CI 2-sided [1.09 to 2.47]
Statistical Analysis 62: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 61]; Test type: Superiority or Other; p = 0.024, ANOVA; LS Mean Difference = 0.56, 95% CI 2-sided [0.07 to 1.04]
Statistical Analysis 63: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 61]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.16, 95% CI 2-sided [0.67 to 1.65]
Statistical Analysis 64: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 61]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.23, 95% CI 2-sided [0.54 to 1.92]
Statistical Analysis 65: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 61]; Test type: Superiority or Other; p = 0.079, ANOVA; LS Mean Difference = 0.62, 95% CI 2-sided [-0.07 to 1.32]
Statistical Analysis 66: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 61]; Test type: Superiority or Other; p = 0.015, ANOVA; LS Mean Difference = 0.60, 95% CI 2-sided [0.12 to 1.09]
Statistical Analysis 67: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 67]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.25, 95% CI 2-sided [0.56 to 1.94]
Statistical Analysis 68: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 67]; Test type: Superiority or Other; p = 0.438, ANOVA; LS Mean Difference = 0.19, 95% CI 2-sided [-0.29 to 0.67]
Statistical Analysis 69: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 67]; Test type: Superiority or Other; p = 0.001, ANOVA; LS Mean Difference = 0.80, 95% CI 2-sided [0.31 to 1.29]
Statistical Analysis 70: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 67]; Test type: Superiority or Other; p = 0.003, ANOVA; LS Mean Difference = 1.06, 95% CI 2-sided [0.37 to 1.75]
Statistical Analysis 71: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 67]; Test type: Superiority or Other; p = 0.204, ANOVA; LS Mean Difference = 0.45, 95% CI 2-sided [-0.25 to 1.14]
Statistical Analysis 72: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 67]; Test type: Superiority or Other; p = 0.014, ANOVA; LS Mean Difference = 0.61, 95% CI 2-sided [0.12 to 1.10]
Statistical Analysis 73: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 73]; Test type: Superiority or Other; p = 0.018, ANOVA; LS Mean Difference = 0.84, 95% CI 2-sided [0.15 to 1.53]
Statistical Analysis 74: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 73]; Test type: Superiority or Other; p = 0.867, ANOVA; LS Mean Difference = 0.04, 95% CI 2-sided [-0.44 to 0.52]
Statistical Analysis 75: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 73]; Test type: Superiority or Other; p = 0.099, ANOVA; LS Mean Difference = 0.41, 95% CI 2-sided [-0.08 to 0.90]
Statistical Analysis 76: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 73]; Test type: Superiority or Other; p = 0.024, ANOVA; LS Mean Difference = 0.80, 95% CI 2-sided [0.11 to 1.49]
Statistical Analysis 77: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 73]; Test type: Superiority or Other; p = 0.228, ANOVA; LS Mean Difference = 0.43, 95% CI 2-sided [-0.27 to 1.12]
Statistical Analysis 78: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 73]; Test type: Superiority or Other; p = 0.136, ANOVA; LS Mean Difference = 0.37, 95% CI 2-sided [-0.12 to 0.86]
Statistical Analysis 79: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 79]; Test type: Superiority or Other; p = 0.078, ANOVA; LS Mean Difference = 0.60, 95% CI 2-sided [-0.07 to 1.28]
Statistical Analysis 80: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 79]; Test type: Superiority or Other; p = 0.716, ANOVA; LS Mean Difference = 0.09, 95% CI 2-sided [-0.38 to 0.56]
Statistical Analysis 81: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 79]; Test type: Superiority or Other; p = 0.197, ANOVA; LS Mean Difference = 0.31, 95% CI 2-sided [-0.16 to 0.79]
Statistical Analysis 82: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 79]; Test type: Superiority or Other; p = 0.131, ANOVA; LS Mean Difference = 0.52, 95% CI 2-sided [-0.15 to 1.19]
Statistical Analysis 83: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 79]; Test type: Superiority or Other; p = 0.399, ANOVA; LS Mean Difference = 0.29, 95% CI 2-sided [-0.39 to 0.97]
Statistical Analysis 84: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 79]; Test type: Superiority or Other; p = 0.349, ANOVA; LS Mean Difference = 0.23, 95% CI 2-sided [-0.25 to 0.70]
Statistical Analysis 85: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 85]; Test type: Superiority or Other; p = 0.169, ANOVA; LS Mean Difference = 0.46, 95% CI 2-sided [-0.20 to 1.12]
Statistical Analysis 86: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 85]; Test type: Superiority or Other; p = 0.937, ANOVA; LS Mean Difference = -0.02, 95% CI 2-sided [-0.48 to 0.44]
Statistical Analysis 87: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 85]; Test type: Superiority or Other; p = 0.351, ANOVA; LS Mean Difference = 0.22, 95% CI 2-sided [-0.25 to 0.69]
Statistical Analysis 88: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 8, analysis 85]; Test type: Superiority or Other; p = 0.151, ANOVA; LS Mean Difference = 0.48, 95% CI 2-sided [-0.18 to 1.14]
Statistical Analysis 89: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 85]; Test type: Superiority or Other; p = 0.476, ANOVA; LS Mean Difference = 0.24, 95% CI 2-sided [-0.42 to 0.90]
Statistical Analysis 90: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 8, analysis 85]; Test type: Superiority or Other; p = 0.310, ANOVA; LS Mean Difference = 0.24, 95% CI 2-sided [-0.22 to 0.71]

12. Other Pre Specified Outcome: Time-weighted Sum of Pain Intensity Difference Scores on 11-Point Numerical Scale (SPID11) From 0 to 2 Hours, 0 to 6 Hours and 0 to 12 Hours Post-dose
Description: Pain intensity was assessed on an 11-point numerical pain severity rating scale. SPID11: Time-weighted sum of PID scores over 12 hours. SPID11 score range was -10 (worst score) to 20 (best score) for SPID 0-2, -30 (worst score) to 60 (best score) for SPID 0-6, -60 (worst score) to 120 (best score) for SPID 0-12. PID was calculated by subtracting the pain intensity score at given post-dose time points (pain severity score range: 0 =no pain to 10 =worst possible pain) from the baseline pain intensity scores (score range: 5 =moderate pain to 10 =worst possible pain; as participants with baseline pain score of at least moderate were included in study). Total possible score range for PID: -5 (worst) to 10 (best).
Time Frame: 0 to 2 hours, 0 to 6 hours, 0 to 12 hours post-dose
Population: FAS included all randomized participants who were dosed with the study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen 250 mg + Acetaminophen 500 mg | Ibuprofen 250 mg | Acetaminophen 650 mg
Number analyzed (Participants) | 56 | 172 | 175 | 165
units on a scale
  0 to 2 hours | 0.3 (2.9) | 7.7 (4.4) | 6.3 (4.6) | 5.7 (4.1)
  0 to 6 hours | 2.9 (13.5) | 27.5 (14.4) | 23.1 (15.6) | 16.0 (14.9)
  0 to 12 hours | 6.8 (30.0) | 41.8 (28.7) | 36.3 (29.3) | 24.7 (29.5)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 0 to 2 hours: Treatment difference and 95% CI were based on LS Mean from ANCOVA with treatment, gender, baseline categorical PSR as classification variables and baseline numerical PSR used as a continuous covariate; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 7.35, 95% CI 2-sided [6.09 to 8.61]
Statistical Analysis 2: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.002, ANCOVA; LS Mean Difference = 1.41, 95% CI 2-sided [0.53 to 2.28]
Statistical Analysis 3: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 1.98, 95% CI 2-sided [1.09 to 2.88]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 5.94, 95% CI 2-sided [4.69 to 7.20]
Statistical Analysis 5: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 5.37, 95% CI 2-sided [4.10 to 6.63]
Statistical Analysis 6: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.203, ANCOVA; LS Mean Difference = 0.58, 95% CI 2-sided [-0.31 to 1.47]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 0 to 6 hours: Treatment difference and 95% CI were based on LS Mean from ANCOVA with treatment, gender, baseline categorical PSR as classification variables and baseline numerical PSR used as a continuous covariate; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 24.50, 95% CI 2-sided [20.10 to 28.90]
Statistical Analysis 8: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 12, analysis 7]; Test type: Superiority or Other; p = 0.005, ANCOVA; LS Mean Difference = 4.44, 95% CI 2-sided [1.37 to 7.52]
Statistical Analysis 9: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 12, analysis 7]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 11.36, 95% CI 2-sided [8.23 to 14.48]
Statistical Analysis 10: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 12, analysis 7]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 20.06, 95% CI 2-sided [15.66 to 24.45]
Statistical Analysis 11: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 12, analysis 7]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 13.14, 95% CI 2-sided [8.71 to 17.57]
Statistical Analysis 12: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 12, analysis 7]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 6.92, 95% CI 2-sided [3.80 to 10.04]
Statistical Analysis 13: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 0 to 12 hours: Treatment difference and 95% CI were based on LS Mean from ANCOVA with treatment, gender, baseline categorical PSR as classification variables and baseline numerical PSR used as a continuous covariate; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 34.83, 95% CI 2-sided [26.09 to 43.57]
Statistical Analysis 14: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 12, analysis 13]; Test type: Superiority or Other; p = 0.060, ANCOVA; LS Mean Difference = 5.85, 95% CI 2-sided [-0.25 to 11.95]
Statistical Analysis 15: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 12, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 16.75, 95% CI 2-sided [10.54 to 22.95]
Statistical Analysis 16: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 12, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 28.98, 95% CI 2-sided [20.26 to 37.71]
Statistical Analysis 17: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 12, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 18.08, 95% CI [9.29 to 26.88]
Statistical Analysis 18: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 12, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 10.90, 95% CI 2-sided [4.70 to 17.10]

13. Other Pre Specified Outcome: Time-weighted Sum of Pain Intensity Difference Scores on 4-Point Categorical Scale (SPID4) From 0 to 2 Hours, 0 to 6 Hours, 0 to 8 Hours, 0 to 12 Hours and 6 to 8 Hours Post-dose
Description: Pain intensity was assessed on a 4-point categorical pain severity rating scale. SPID4: Time-weighted sum of PID over post-dose time points. SPID4 score range was -2 (worst score) to 6 (best score) for SPID 0-2, -6 (worst score) to 18 (best score) for SPID 0-6, -8 (worst score) to 24 (best score) for SPID 0-8, -12 (worst score) to 36 (best score) for SPID 0-12 and -3 (worst score) to 9 (best score) for SPID 6-8. PID was calculated by subtracting the pain intensity score at given post-dose time points (pain severity score range: 0 [none] to 3 [severe]) from the baseline pain intensity scores (score range: 2 =moderate pain to 3 = severe pain; as participants with baseline pain score of at least moderate were included in study). Total possible score range for PID: -1 (worst score) to 3 (best score).
Time Frame: 0 to 2 hours, 0 to 6 hours, 0 to 8 hours, 0 to 12, 6 to 8 hours post-dose
Population: FAS included all randomized participants who were dosed with the study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen 250 mg + Acetaminophen 500 mg | Ibuprofen 250 mg | Acetaminophen 650 mg
Number analyzed (Participants) | 56 | 172 | 175 | 165
units on a scale
  0 to 2 hours | 0.1 (0.9) | 2.2 (1.5) | 1.7 (1.7) | 1.6 (1.4)
  0 to 6 hours | 0.7 (4.2) | 8.0 (4.9) | 6.4 (5.5) | 4.6 (4.7)
  0 to 8 hours | 0.9 (5.8) | 9.9 (6.6) | 7.9 (7.1) | 5.5 (6.2)
  0 to 12 hours | 1.4 (9.0) | 11.9 (9.6) | 9.8 (9.9) | 6.8 (9.0)
  6 to 8 hours | 0.4 (2.6) | 3.2 (3.0) | 2.5 (2.9) | 1.6 (2.7)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 0-2 hour: Treatment difference and 95% CI were based on LS Mean from ANOVA with treatment, gender and baseline categorical PSR; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 2.12, 95% CI 2-sided [1.72 to 2.51]
Statistical Analysis 2: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.002, ANOVA; LS Mean Difference = 0.44, 95% CI 2-sided [0.16 to 0.71]
Statistical Analysis 3: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.58, 95% CI 2-sided [0.30 to 0.86]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.68, 95% CI 2-sided [1.29 to 2.08]
Statistical Analysis 5: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.53, 95% CI 2-sided [1.14 to 1.93]
Statistical Analysis 6: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.303, ANOVA; LS Mean Difference = 0.15, 95% CI 2-sided [-0.13 to 0.43]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 0-6 hour: Treatment difference and 95% CI were based on LS Mean from ANOVA with treatment, gender and baseline categorical PSR; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 7.22, 95% CI 2-sided [5.86 to 8.58]
Statistical Analysis 8: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 13, analysis 7]; Test type: Superiority or Other; p = 0.001, ANOVA; LS Mean Difference = 1.58, 95% CI 2-sided [0.63 to 2.53]
Statistical Analysis 9: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 13, analysis 7]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 3.48, 95% CI 2-sided [2.52 to 4.45]
Statistical Analysis 10: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 13, analysis 7]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 5.64, 95% CI 2-sided [4.28 to 6.99]
Statistical Analysis 11: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 13, analysis 7]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 3.73, 95% CI 2-sided [2.37 to 5.10]
Statistical Analysis 12: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 13, analysis 7]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.90, 95% CI 2-sided [0.95 to 2.86]
Statistical Analysis 13: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 0-8 hour: Treatment difference and 95% CI were based on LS Mean from ANOVA with treatment, gender and baseline categorical PSR; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 8.89, 95% CI 2-sided [7.08 to 10.71]
Statistical Analysis 14: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 13, analysis 13]; Test type: Superiority or Other; p = 0.002, ANOVA; LS Mean Difference = 2.00, 95% CI 2-sided [0.73 to 3.26]
Statistical Analysis 15: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 13, analysis 13]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 4.48, 95% CI 2-sided [3.20 to 5.77]
Statistical Analysis 16: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 13, analysis 13]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 6.90, 95% CI 2-sided [5.08 to 8.71]
Statistical Analysis 17: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 13, analysis 13]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 4.41, 95% CI 2-sided [2.58 to 6.24]
Statistical Analysis 18: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 13, analysis 13]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 2.49, 95% CI 2-sided [1.21 to 3.77]
Statistical Analysis 19: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 0-12 hour: Treatment difference and 95% CI were based on LS Mean from ANOVA with treatment, gender and baseline categorical PSR; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 10.42, 95% CI 2-sided [7.76 to 13.08]
Statistical Analysis 20: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 13, analysis 19]; Test type: Superiority or Other; p = 0.024, ANOVA; LS Mean Difference = 2.14, 95% CI 2-sided [0.28 to 4.00]
Statistical Analysis 21: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 13, analysis 19]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 5.24, 95% CI 2-sided [3.35 to 7.12]
Statistical Analysis 22: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 13, analysis 19]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 8.28, 95% CI 2-sided [5.62 to 10.93]
Statistical Analysis 23: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 13, analysis 19]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 5.18, 95% CI 2-sided [2.51 to 7.86]
Statistical Analysis 24: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 13, analysis 19]; Test type: Superiority or Other; p = 0.001, ANOVA; LS Mean Difference = 3.10, 95% CI 2-sided [1.22 to 4.97]
Statistical Analysis 25: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 6-8 hour: Treatment difference and 95% CI were based on LS Mean from ANOVA with treatment, gender and baseline categorical PSR; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 2.77, 95% CI 2-sided [1.95 to 3.59]
Statistical Analysis 26: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 13, analysis 25]; Test type: Superiority or Other; p = 0.023, ANOVA; LS Mean Difference = 0.66, 95% CI 2-sided [0.09 to 1.24]
Statistical Analysis 27: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 13, analysis 25]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.66, 95% CI 2-sided [1.07 to 2.24]
Statistical Analysis 28: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 13, analysis 25]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 2.11, 95% CI 2-sided [1.29 to 2.92]
Statistical Analysis 29: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 13, analysis 25]; Test type: Superiority or Other; p = 0.008, ANOVA; LS Mean Difference = 1.11, 95% CI 2-sided [0.29 to 1.94]
Statistical Analysis 30: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 13, analysis 25]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.99, 95% CI 2-sided [0.41 to 1.57]

14. Other Pre Specified Outcome: Time-weighted Sum of Pain Relief Rating (TOTPAR) From 0 to 2 Hours, 0 to 6 Hours and 0 to 12 Hours Post Dose
Description: TOTPAR: Time-weighted sum of PRR scores over 2, 6 and 12 hours. TOTPAR total score range: 0 (worst score) to 8 (best score) for TOTPAR 0-2, 0 (worst score) to 24 (best score) for TOTPAR 0-6, 0 (worst score) to 32 (best score) for TOTPAR 0-8, 0 (worst score) to 48 (best score) for TOTPAR 0-12. PRR was assessed on a 5-point categorical pain relief rating scale which ranges from 0 =no relief to 4 =complete relief.
Time Frame: 0 to 2 hours, 0 to 6 hours, 0 to 12 hours post-dose
Population: FAS included all randomized participants who were dosed with the study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen 250 mg + Acetaminophen 500 mg | Ibuprofen 250 mg | Acetaminophen 650 mg
Number analyzed (Participants) | 56 | 172 | 175 | 165
units on a scale
  0 to 2 hours | 0.9 (1.2) | 4.1 (2.0) | 3.5 (2.0) | 3.2 (1.9)
  0 to 6 hours | 3.8 (5.6) | 14.6 (6.3) | 12.3 (6.8) | 9.2 (6.7)
  0 to 12 hours | 8.3 (12.7) | 23.0 (12.7) | 19.9 (13.2) | 15.0 (13.4)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 0 to 2 hours: Treatment difference and 95% CI were based on LS Mean from ANOVA with treatment, gender and baseline categorical PSR; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 3.25, 95% CI 2-sided [2.68 to 3.82]
Statistical Analysis 2: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; 0-2 hour:Treatment difference and 95% CI were based on LS Mean from ANOVA with treatment, gender and baseline categorical PSR; Test type: Superiority or Other; p = 0.002, ANOVA; LS Mean Difference = 0.63, 95% CI 2-sided [0.23 to 1.03]
Statistical Analysis 3: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.86, 95% CI 2-sided [0.46 to 1.27]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 2.62, 95% CI 2-sided [2.05 to 3.19]
Statistical Analysis 5: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 2.39, 95% CI 2-sided [1.81 to 2.96]
Statistical Analysis 6: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.258, ANOVA; LS Mean Difference = 0.23, 95% CI 2-sided [-0.17 to 0.64]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 0 to 6 hours: Treatment difference and 95% CI were based on LS Mean from ANOVA with treatment, gender and baseline categorical PSR; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 10.77, 95% CI 2-sided [8.79 to 12.74]
Statistical Analysis 8: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p = 0.001, ANOVA; LS Mean Difference = 2.29, 95% CI 2-sided [0.91 to 3.67]
Statistical Analysis 9: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 5.33, 95% CI 2-sided [3.93 to 6.73]
Statistical Analysis 10: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 8.48, 95% CI 2-sided [6.51 to 10.44]
Statistical Analysis 11: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 5.44, 95% CI 2-sided [3.46 to 7.42]
Statistical Analysis 12: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 3.04, 95% CI 2-sided [1.65 to 4.43]
Statistical Analysis 13: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 0 to 12 hours: Treatment difference and 95% CI were based on LS Mean from ANOVA with treatment, gender and baseline categorical PSR; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 14.68, 95% CI 2-sided [10.74 to 18.62]
Statistical Analysis 14: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p = 0.024, ANOVA; LS Mean Difference = 3.16, 95% CI 2-sided [0.41 to 5.91]
Statistical Analysis 15: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 7.94, 95% CI 2-sided [5.15 to 10.73]
Statistical Analysis 16: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 11.52, 95% CI 2-sided [7.59 to 15.45]
Statistical Analysis 17: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 6.75, 95% CI [2.79 to 10.71]
Statistical Analysis 18: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 4.78, 95% CI 2-sided [2.0 to 7.56]

15. Other Pre Specified Outcome: Time-weighted Sum of Pain Relief Rating and Pain Intensity Difference Scores on 4-Point Categorical Scale (SPRID4) Over 2, 6, 8, 12 and 6 to 8 Hours Post-dose
Description: SPRID4: Time-weighted sum of PRR and PID based on 4 point categorical pain severity rating scale (PRID) with score range: -2(worst score) to 14 (best score) for SPRID 0-2, -6 (worst score) to 42 (best score) for SPRID 0-6, -8 (worst score) to 56 (best score) for SPRID 0-8, -12 (worst score) to 84 (best score) for SPRID 0-12 and -3 (worst score) to 21 (best score) for SPRID 6-8 hours. PRID: sum of PID and PRR at post-dose time point with score range: -1 (worst score) to 7 (best score). PID calculated by subtracting pain intensity score at post-dose time points (score range: 0 [none] to 3 [severe]) from baseline pain intensity scores (score range: 2 =moderate pain to 3 = severe pain; as participants with baseline score of at least moderate were included). PID total possible score range: -1 (worst score) to 3(best score). PRR assessed on 5-point categorical scale with range: 0 =no relief to 4 =complete relief.
Time Frame: 0 to 2 hours, 0 to 6 hours, 0 to 8 hours, 0 to 12, 6 to 8 hours post-dose
Population: FAS included all randomized participants who were dosed with the study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen 250 mg + Acetaminophen 500 mg | Ibuprofen 250 mg | Acetaminophen 650 mg
Number analyzed (Participants) | 56 | 172 | 175 | 165
units on a scale
  0 to 2 hours | 0.9 (2.0) | 6.3 (3.3) | 5.2 (3.5) | 4.9 (3.1)
  0 to 6 hours | 4.5 (9.3) | 22.5 (10.7) | 18.6 (11.9) | 13.8 (11.0)
  0 to 8 hours | 6.2 (13.0) | 28.2 (14.5) | 23.2 (15.7) | 16.9 (14.8)
  0 to 12 hours | 9.7 (20.5) | 34.9 (21.5) | 29.6 (22.5) | 21.9 (21.6)
  6 to 8 hours | 2.7 (6.1) | 9.3 (6.9) | 7.6 (6.7) | 5.0 (6.6)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 5.37, 95% CI 2-sided [4.42 to 6.32]
Statistical Analysis 2: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.002, ANOVA; LS Mean Difference = 1.07, 95% CI 2-sided [0.40 to 1.74]
Statistical Analysis 3: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 1.45, 95% CI 2-sided [0.77 to 2.13]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 4.30, 95% CI 2-sided [3.35 to 5.25]
Statistical Analysis 5: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 3.92, 95% CI 2-sided [2.96 to 4.88]
Statistical Analysis 6: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.268, ANOVA; LS Mean Difference = 0.38, 95% CI 2-sided [-0.29 to 1.05]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 13, analysis 7]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 17.99, 95% CI 2-sided [14.69 to 21.28]
Statistical Analysis 8: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 13, analysis 7]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 3.87, 95% CI 2-sided [1.57 to 6.17]
Statistical Analysis 9: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 13, analysis 7]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 8.81, 95% CI 2-sided [6.48 to 11.15]
Statistical Analysis 10: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 13, analysis 7]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 14.12, 95% CI 2-sided [10.83 to 17.40]
Statistical Analysis 11: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 13, analysis 7]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 9.17, 95% CI 2-sided [5.86 to 12.48]
Statistical Analysis 12: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 13, analysis 7]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 4.94, 95% CI 2-sided [2.62 to 7.27]
Statistical Analysis 13: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 13, analysis 13]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 21.94, 95% CI 2-sided [17.52 to 26.37]
Statistical Analysis 14: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 13, analysis 13]; Test type: Superiority or Other; p = 0.002, ANOVA; LS Mean Difference = 5.00, 95% CI 2-sided [1.91 to 8.09]
Statistical Analysis 15: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 13, analysis 13]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 11.43, 95% CI 2-sided [8.29 to 14.56]
Statistical Analysis 16: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 13, analysis 13]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 16.94, 95% CI 2-sided [12.53 to 21.36]
Statistical Analysis 17: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 13, analysis 13]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 10.52, 95% CI 2-sided [6.07 to 14.97]
Statistical Analysis 18: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 13, analysis 13]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 6.43, 95% CI 2-sided [3.30 to 9.55]
Statistical Analysis 19: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 13, analysis 19]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 25.10, 95% CI 2-sided [18.57 to 31.63]
Statistical Analysis 20: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 13, analysis 19]; Test type: Superiority or Other; p = 0.023, ANOVA; LS Mean Difference = 5.30, 95% CI 2-sided [0.74 to 9.86]
Statistical Analysis 21: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 13, analysis 19]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 13.17, 95% CI 2-sided [8.55 to 17.80]
Statistical Analysis 22: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 13, analysis 19]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 19.80, 95% CI 2-sided [13.28 to 26.31]
Statistical Analysis 23: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 13, analysis 19]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 11.93, 95% CI 2-sided [5.36 to 18.49]
Statistical Analysis 24: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 13, analysis 19]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 7.87, 95% CI 2-sided [3.27 to 12.48]
Statistical Analysis 25: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 13, analysis 25]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 6.61, 95% CI 2-sided [4.61 to 8.62]
Statistical Analysis 26: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 13, analysis 25]; Test type: Superiority or Other; p = 0.015, ANOVA; LS Mean Difference = 1.74, 95% CI 2-sided [0.34 to 3.14]
Statistical Analysis 27: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 13, analysis 25]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 4.34, 95% CI 2-sided [2.92 to 5.76]
Statistical Analysis 28: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 13, analysis 25]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 4.87, 95% CI 2-sided [2.87 to 6.88]
Statistical Analysis 29: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 13, analysis 25]; Test type: Superiority or Other; p = 0.028, ANOVA; LS Mean Difference = 2.27, 95% CI 2-sided [0.25 to 4.28]
Statistical Analysis 30: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 13, analysis 25]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 2.61, 95% CI 2-sided [1.19 to 4.02]

16. Other Pre Specified Outcome: Cumulative Percentage of Participants With Treatment Failure
Description: as for outcome 5
Time Frame: 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 hours post-dose
Population: FAS included all randomized participants who were dosed with the study medication and provided a baseline assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ibuprofen 250 mg + Acetaminophen 500 mg | Ibuprofen 250 mg | Acetaminophen 650 mg
Number analyzed (Participants) | 56 | 172 | 175 | 165
percentage of participants
  1.5 hour | 39.3 | 2.9 | 6.9 | 6.7
  2 hour | 51.8 | 4.1 | 10.3 | 10.3
  3 hour | 62.5 | 7.0 | 13.1 | 18.8
  4 hour | 64.3 | 7.6 | 16.6 | 27.9
  5 hour | 66.1 | 8.1 | 18.3 | 35.2
  6 hour | 67.9 | 10.5 | 21.7 | 38.8
  7 hour | 69.6 | 16.9 | 25.7 | 44.2
  8 hour | 69.6 | 24.4 | 33.1 | 51.5
  9 hour | 69.6 | 35.5 | 42.3 | 56.4
  10 hour | 69.6 | 46.5 | 48.6 | 60.0
  11 hour | 69.6 | 51.7 | 55.4 | 62.4
  12 hour | 71.4 | 55.8 | 60.0 | 63.6
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 1.5 hour: Treatment difference and its associated 95% CI were calculated based on CMH adjusted proportions and the corresponding standard errors, controlling for baseline categorical PSR and gender using table scores; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -36.56, 95% CI 2-sided [-49.41 to -23.71]
Statistical Analysis 2: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; p = 0.086, Cochran-Mantel-Haenszel; CMH adjusted proportions = -3.95, 95% CI 2-sided [-8.45 to 0.56]
Statistical Analysis 3: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; p = 0.112, Cochran-Mantel-Haenszel; CMH adjusted proportions = -3.71, 95% CI 2-sided [-8.28 to 0.86]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -32.52, 95% CI 2-sided [-45.86 to -19.17]
Statistical Analysis 5: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -32.88, 95% CI 2-sided [-46.22 to -19.55]
Statistical Analysis 6: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; p = 0.968, Cochran-Mantel-Haenszel; CMH adjusted proportions = 0.11, 95% CI 2-sided [-5.20 to 5.42]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 2 hour: Treatment difference and its associated 95% CI were calculated based on CMH adjusted proportions and the corresponding standard errors, controlling for baseline categorical PSR and gender using table scores; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -47.88, 95% CI 2-sided [-61.18 to -34.58]
Statistical Analysis 8: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 7]; Test type: Superiority or Other; p = 0.023, Cochran-Mantel-Haenszel; CMH adjusted proportions = -6.23, 95% CI 2-sided [-11.61 to -0.84]
Statistical Analysis 9: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 7]; Test type: Superiority or Other; p = 0.026, Cochran-Mantel-Haenszel; CMH adjusted proportions = -6.23, 95% CI 2-sided [-11.73 to -0.73]
Statistical Analysis 10: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 7]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -41.51, 95% CI 2-sided [-55.51 to -27.52]
Statistical Analysis 11: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 7]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -41.77, 95% CI 2-sided [-55.65 to -27.89]
Statistical Analysis 12: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 7]; Test type: Superiority or Other; p = 0.960, Cochran-Mantel-Haenszel; CMH adjusted proportions = -0.16, 95% CI 2-sided [-6.56 to 6.23]
Statistical Analysis 13: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 3 hour: Treatment difference and its associated 95% CI were calculated based on CMH adjusted proportions and the corresponding standard errors, controlling for baseline categorical PSR and gender using table scores; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -55.73, 95% CI 2-sided [-68.81 to -42.65]
Statistical Analysis 14: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 13]; Test type: Superiority or Other; p = 0.055, Cochran-Mantel-Haenszel; CMH adjusted proportions = -6.16, 95% CI 2-sided [-12.46 to 0.13]
Statistical Analysis 15: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 13]; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -11.70, 95% CI 2-sided [-18.70 to -4.70]
Statistical Analysis 16: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 13]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -49.41, 95% CI 2-sided [-63.21 to -35.60]
Statistical Analysis 17: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 13]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -44.30, 95% CI 2-sided [-58.04 to -30.55]
Statistical Analysis 18: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 13]; Test type: Superiority or Other; p = 0.151, Cochran-Mantel-Haenszel; CMH adjusted proportions = -5.69, 95% CI 2-sided [-13.46 to 2.08]
Statistical Analysis 19: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 4 hour: Treatment difference and its associated 95% CI were calculated based on CMH adjusted proportions and the corresponding standard errors, controlling for baseline categorical PSR and gender using table scores; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -56.94, 95% CI 2-sided [-69.96 to -43.91]
Statistical Analysis 20: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 19]; Test type: Superiority or Other; p = 0.010, Cochran-Mantel-Haenszel; CMH adjusted proportions = -9.00, 95% CI 2-sided [-15.80 to -2.19]
Statistical Analysis 21: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 19]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -20.11, 95% CI 2-sided [-27.97 to -12.24]
Statistical Analysis 22: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 19]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -47.73, 95% CI 2-sided [-61.64 to -33.83]
Statistical Analysis 23: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 19]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -37.18, 95% CI 2-sided [-50.96 to -23.40]
Statistical Analysis 24: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 19]; Test type: Superiority or Other; p = 0.013, Cochran-Mantel-Haenszel; CMH adjusted proportions = -11.19, 95% CI 2-sided [-20.02 to -2.36]
Statistical Analysis 25: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 5 hour: Treatment difference and its associated 95% CI were calculated based on CMH adjusted proportions and the corresponding standard errors, controlling for baseline categorical PSR and gender using table scores; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -58.14, 95% CI 2-sided [-71.03 to -45.26]
Statistical Analysis 26: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 25]; Test type: Superiority or Other; p = 0.005, Cochran-Mantel-Haenszel; CMH adjusted proportions = -10.15, 95% CI 2-sided [-17.24 to -3.06]
Statistical Analysis 27: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 25]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -26.77, 95% CI 2-sided [-35.10 to -18.44]
Statistical Analysis 28: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 25]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -47.74, 95% CI 2-sided [-61.76 to -33.72]
Statistical Analysis 29: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 25]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -31.69, 95% CI 2-sided [-45.61 to -17.76]
Statistical Analysis 30: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 25]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -16.76, 95% CI 2-sided [-26.10 to -7.42]
Statistical Analysis 31: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 6 hour: Treatment difference and its associated 95% CI were calculated based on CMH adjusted proportions and the corresponding standard errors, controlling for baseline categorical PSR and gender using table scores; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -57.58, 95% CI 2-sided [-70.44 to -44.72]
Statistical Analysis 32: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 31]; Test type: Superiority or Other; p = 0.004, Cochran-Mantel-Haenszel; CMH adjusted proportions = -11.28, 95% CI 2-sided [-18.99 to -3.57]
Statistical Analysis 33: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 31]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -28.06, 95% CI 2-sided [-36.77 to -19.35]
Statistical Analysis 34: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 31]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -46.01, 95% CI 2-sided [-59.98 to -32.04]
Statistical Analysis 35: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 31]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -29.70, 95% CI 2-sided [-43.65 to -15.75]
Statistical Analysis 36: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 31]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -16.94, 95% CI 2-sided [-26.59 to -7.29]
Statistical Analysis 37: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 7 hour: Treatment difference and its associated 95% CI were calculated based on CMH adjusted proportions and the corresponding standard errors, controlling for baseline categorical PSR and gender using table scores; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -52.90, 95% CI 2-sided [-66.06 to -39.75]
Statistical Analysis 38: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 37]; Test type: Superiority or Other; p = 0.042, Cochran-Mantel-Haenszel; CMH adjusted proportions = -8.93, 95% CI 2-sided [-17.53 to -0.34]
Statistical Analysis 39: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 37]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -27.25, 95% CI 2-sided [-36.65 to -17.86]
Statistical Analysis 40: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 37]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -43.78, 95% CI 2-sided [-57.83 to -29.72]
Statistical Analysis 41: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 37]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -25.75, 95% CI 2-sided [-39.93 to -11.57]
Statistical Analysis 42: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 37]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -18.49, 95% CI 2-sided [-28.39 to -8.59]
Statistical Analysis 43: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 8 hour: Treatment difference and its associated 95% CI were calculated based on CMH adjusted proportions and the corresponding standard errors, controlling for baseline categorical PSR and gender using table scores; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -45.27, 95% CI 2-sided [-58.96 to -31.58]
Statistical Analysis 44: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 43]; Test type: Superiority or Other; p = 0.064, Cochran-Mantel-Haenszel; CMH adjusted proportions = -8.88, 95% CI 2-sided [-18.27 to 0.50]
Statistical Analysis 45: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 43]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -26.98, 95% CI 2-sided [-36.91 to -17.05]
Statistical Analysis 46: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 43]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -36.26, 95% CI 2-sided [-50.45 to -22.07]
Statistical Analysis 47: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 43]; Test type: Superiority or Other; p = 0.010, Cochran-Mantel-Haenszel; CMH adjusted proportions = -18.58, 95% CI 2-sided [-32.64 to -4.52]
Statistical Analysis 48: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 43]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -18.17, 95% CI 2-sided [-28.44 to -7.90]
Statistical Analysis 49: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 9 hour: Treatment difference and its associated 95% CI were calculated based on CMH adjusted proportions and the corresponding standard errors, controlling for baseline categorical PSR and gender using table scores; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -34.21, 95% CI 2-sided [-48.21 to -20.21]
Statistical Analysis 50: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 49]; Test type: Superiority or Other; p = 0.179, Cochran-Mantel-Haenszel; CMH adjusted proportions = -6.97, 95% CI 2-sided [-17.12 to 3.19]
Statistical Analysis 51: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 49]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -20.70, 95% CI 2-sided [-31.04 to -10.35]
Statistical Analysis 52: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 49]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -27.20, 95% CI 2-sided [-41.44 to -12.96]
Statistical Analysis 53: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 49]; Test type: Superiority or Other; p = 0.051, Cochran-Mantel-Haenszel; CMH adjusted proportions = -13.90, 95% CI 2-sided [-27.84 to 0.04]
Statistical Analysis 54: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 49]; Test type: Superiority or Other; p = 0.010, Cochran-Mantel-Haenszel; CMH adjusted proportions = -13.76, 95% CI 2-sided [-24.21 to -3.31]
Statistical Analysis 55: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 10 hour: Treatment difference and its associated 95% CI were calculated based on CMH adjusted proportions and the corresponding standard errors, controlling for baseline categorical PSR and gender using table scores; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = -23.25, 95% CI 2-sided [-37.31 to -9.20]
Statistical Analysis 56: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 55]; Test type: Superiority or Other; p = 0.676, Cochran-Mantel-Haenszel; CMH adjusted proportions = -2.22, 95% CI 2-sided [-12.63 to 8.19]
Statistical Analysis 57: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 55]; Test type: Superiority or Other; p = 0.013, Cochran-Mantel-Haenszel; CMH adjusted proportions = -13.15, 95% CI 2-sided [-23.57 to -2.74]
Statistical Analysis 58: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 55]; Test type: Superiority or Other; p = 0.004, Cochran-Mantel-Haenszel; CMH adjusted proportions = -20.94, 95% CI 2-sided [-35.18 to -6.69]
Statistical Analysis 59: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 55]; Test type: Superiority or Other; p = 0.140, Cochran-Mantel-Haenszel; CMH adjusted proportions = -10.39, 95% CI 2-sided [-24.19 to 3.40]
Statistical Analysis 60: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 55]; Test type: Superiority or Other; p = 0.038, Cochran-Mantel-Haenszel; CMH adjusted proportions = -11.06, 95% CI 2-sided [-21.51 to -0.61]
Statistical Analysis 61: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 11 hour: Treatment difference and its associated 95% CI were calculated based on CMH adjusted proportions and the corresponding standard errors, controlling for baseline categorical PSR and gender using table scores; Test type: Superiority or Other; p = 0.013, Cochran-Mantel-Haenszel; CMH adjusted proportions = -17.9, 95% CI [-32.13 to -3.79]
Statistical Analysis 62: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 61]; Test type: Superiority or Other; p = 0.467, Cochran-Mantel-Haenszel; CMH adjusted proportions = -3.85, 95% CI [-14.23 to 6.53]
Statistical Analysis 63: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 61]; Test type: Superiority or Other; p = 0.049, Cochran-Mantel-Haenszel; CMH adjusted proportions = -10.38, 95% CI [-20.73 to -0.02]
Statistical Analysis 64: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 61]; Test type: Superiority or Other; p = 0.050, Cochran-Mantel-Haenszel; CMH adjusted proportions = -14.10, 95% CI [-28.22 to 0.02]
Statistical Analysis 65: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 61]; Test type: Superiority or Other; p = 0.255, Cochran-Mantel-Haenszel; CMH adjusted proportions = -7.99, 95% CI [-21.73 to 5.76]
Statistical Analysis 66: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 61]; Test type: Superiority or Other; p = 0.212, Cochran-Mantel-Haenszel; CMH adjusted proportions = -6.57, 95% CI [-16.89 to 3.75]
Statistical Analysis 67: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 12 hour: Treatment difference and its associated 95% CI were calculated based on CMH adjusted proportions and the corresponding standard errors, controlling for baseline categorical PSR and gender using table scores; Test type: Superiority or Other; p = 0.027, Cochran-Mantel-Haenszel; CMH adjusted proportions = -15.68, 95% CI [-29.59 to -1.77]
Statistical Analysis 68: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 67]; Test type: Superiority or Other; p = 0.399, Cochran-Mantel-Haenszel; CMH adjusted proportions = -4.39, 95% CI 2-sided [-14.59 to 5.82]
Statistical Analysis 69: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 67]; Test type: Superiority or Other; p = 0.152, Cochran-Mantel-Haenszel; CMH adjusted proportions = -7.50, 95% CI [-17.76 to 2.77]
Statistical Analysis 70: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 67]; Test type: Superiority or Other; p = 0.106, Cochran-Mantel-Haenszel; CMH adjusted proportions = -11.32, 95% CI 2-sided [-25.05 to 2.40]
Statistical Analysis 71: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 67]; Test type: Superiority or Other; p = 0.210, Cochran-Mantel-Haenszel; CMH adjusted proportions = -8.59, 95% CI [-22.00 to 4.83]
Statistical Analysis 72: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 67]; Test type: Superiority or Other; p = 0.545, Cochran-Mantel-Haenszel; CMH adjusted proportions = -3.13, 95% CI [-13.26 to 7.00]

17. Other Pre Specified Outcome: Cumulative Percentage of Participants With Confirmed First Perceptible Relief
Description: Percentage of participants with confirmed first perceptible relief was reported. Participants evaluated the time to first perceptible relief (confirmed by meaningful relief) by stopping the first stopwatch labelled 'first perceptible relief' at the moment they first began to experience any pain relief, if the participant also achieved meaningful relief by the end of the study. Stopwatch was active up to 12 hours after dosing or until stopped by the participant, or until the participant dropped out due to treatment failure prior to depressing the first stopwatch or until the time of withdrawal (discontinuation). Treatment failure was defined as participant taking rescue medication, or discontinuing due to lack of efficacy.
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 hours post-dose
Population: FAS included all randomized participants who were dosed with the study medication and provided a baseline assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ibuprofen 250 mg + Acetaminophen 500 mg | Ibuprofen 250 mg | Acetaminophen 650 mg
Number analyzed (Participants) | 56 | 172 | 175 | 165
percentage of participants
  0.25 hour | 8.9 | 29.7 | 25.1 | 26.1
  0.5 hour | 16.1 | 66.9 | 61.7 | 57.0
  1 hour | 21.4 | 81.4 | 77.1 | 71.5
  1.5 hour | 25.0 | 84.9 | 79.4 | 71.5
  2 hour | 25.0 | 85.5 | 79.4 | 71.5
  3 hour | 28.6 | 86.6 | 79.4 | 71.5
  4 hour | 28.6 | 86.6 | 79.4 | 71.5
  5 hour | 28.6 | 86.6 | 79.4 | 71.5
  6 hour | 28.6 | 86.6 | 79.4 | 71.5
  7 hour | 28.6 | 86.6 | 79.4 | 71.5
  8 hour | 28.6 | 86.6 | 79.4 | 71.5
  9 hour | 28.6 | 86.6 | 79.4 | 71.5
  10 hour | 28.6 | 86.6 | 79.4 | 71.5
  11 hour | 28.6 | 86.6 | 79.4 | 71.5
  12 hour | 28.6 | 86.6 | 79.4 | 71.5
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 0.25 hour: Treatment difference and its associated 95% CI were calculated based on CMH adjusted proportions and the corresponding standard errors, controlling for baseline categorical PSR and gender using table scores; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 20.74, 95% CI 2-sided [10.54 to 30.94]
Statistical Analysis 2: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; p = 0.342, Cochran-Mantel-Haenszel; CMH adjusted proportions = 4.52, 95% CI 2-sided [-4.81 to 13.86]
Statistical Analysis 3: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; p = 0.459, Cochran-Mantel-Haenszel; CMH adjusted proportions = 3.62, 95% CI 2-sided [-5.98 to 13.22]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 16.20, 95% CI 2-sided [6.24 to 26.17]
Statistical Analysis 5: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 17.37, 95% CI 2-sided [7.42 to 27.31]
Statistical Analysis 6: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; p = 0.849, Cochran-Mantel-Haenszel; CMH adjusted proportions = -0.91, 95% CI 2-sided [-10.2 to 8.42]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 0.5 hour: Treatment difference and its associated 95% CI were calculated based on CMH adjusted proportions and the corresponding standard errors, controlling for baseline categorical PSR and gender using table scores; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 51.08, 95% CI 2-sided [39.53 to 62.62]
Statistical Analysis 8: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 17, analysis 7]; Test type: Superiority or Other; p = 0.318, Cochran-Mantel-Haenszel; Cumulative Percentage of Participants wi = 5.16, 95% CI 2-sided [-4.97 to 15.30]
Statistical Analysis 9: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 17, analysis 7]; Test type: Superiority or Other; p = 0.062, Cochran-Mantel-Haenszel; CMH adjusted proportions = 9.86, 95% CI 2-sided [-0.49 to 20.21]
Statistical Analysis 10: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 17, analysis 7]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 45.60, 95% CI 2-sided [33.45 to 57.76]
Statistical Analysis 11: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 17, analysis 7]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 41.07, 95% CI 2-sided [28.76 to 53.38]
Statistical Analysis 12: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 17, analysis 7]; Test type: Superiority or Other; p = 0.374, Cochran-Mantel-Haenszel; CMH adjusted proportions = 4.74, 95% CI 2-sided [-5.70 to 15.17]
Statistical Analysis 13: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 1 hour: Treatment difference and its associated 95% CI were calculated based on CMH adjusted proportions and the corresponding standard errors, controlling for baseline categorical PSR and gender using table scores; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 60.09, 95% CI 2-sided [47.93 to 72.26]
Statistical Analysis 14: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 17, analysis 13]; Test type: Superiority or Other; p = 0.323, Cochran-Mantel-Haenszel; CMH adjusted proportions = 4.30, 95% CI 2-sided [-4.22 to 12.81]
Statistical Analysis 15: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 17, analysis 13]; Test type: Superiority or Other; p = 0.032, Cochran-Mantel-Haenszel; CMH adjusted proportions = 9.86, 95% CI 2-sided [0.86 to 18.86]
Statistical Analysis 16: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 17, analysis 13]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 55.66, 95% CI 2-sided [43.11 to 68.20]
Statistical Analysis 17: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 17, analysis 13]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 50.38, 95% CI 2-sided [37.71 to 63.05]
Statistical Analysis 18: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 17, analysis 13]; Test type: Superiority or Other; p = 0.232, Cochran-Mantel-Haenszel; CMH adjusted proportions = 5.61, 95% CI 2-sided [-3.58 to 14.80]
Statistical Analysis 19: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 59.92, 95% CI 2-sided [47.39 to 72.46]
Statistical Analysis 20: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; p = 0.179, Cochran-Mantel-Haenszel; CMH adjusted proportions = 5.51, 95% CI 2-sided [-2.52 to 13.53]
Statistical Analysis 21: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; p = 0.003, Cochran-Mantel-Haenszel; CMH adjusted proportions = 13.37, 95% CI 2-sided [4.65 to 22.10]
Statistical Analysis 22: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 54.32, 95% CI 2-sided [41.36 to 67.29]
Statistical Analysis 23: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 46.74, 95% CI 2-sided [33.50 to 59.99]
Statistical Analysis 24: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; p = 0.087, Cochran-Mantel-Haenszel; CMH adjusted proportions = 7.91, 95% CI 2-sided [-1.15 to 16.97]
Statistical Analysis 25: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 16, analysis 7]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 60.51, 95% CI 2-sided [47.99 to 73.03]
Statistical Analysis 26: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 7]; Test type: Superiority or Other; p = 0.135, Cochran-Mantel-Haenszel; CMH adjusted proportions = 6.08, 95% CI 2-sided [-1.89 to 14.05]
Statistical Analysis 27: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 7]; Test type: Superiority or Other; p = 0.002, Cochran-Mantel-Haenszel; CMH adjusted proportions = 13.97, 95% CI 2-sided [5.30 to 22.64]
Statistical Analysis 28: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 7]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 54.32, 95% CI 2-sided [41.36 to 67.29]
Statistical Analysis 29: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 7]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 46.74, 95% CI 2-sided [33.50 to 59.99]
Statistical Analysis 30: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 7]; Test type: Superiority or Other; p = 0.087, Cochran-Mantel-Haenszel; CMH adjusted proportions = 7.91, 95% CI 2-sided [-1.15 to 16.97]
Statistical Analysis 31: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 16, analysis 13]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 58.12, 95% CI 2-sided [45.24 to 71.00]
Statistical Analysis 32: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 13]; Test type: Superiority or Other; p = 0.071, Cochran-Mantel-Haenszel; CMH adjusted proportions = 7.23, 95% CI 2-sided [-0.63 to 15.10]
Statistical Analysis 33: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 13]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 15.12, 95% CI 2-sided [6.55 to 23.69]
Statistical Analysis 34: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 13]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 50.74, 95% CI 2-sided [37.39 to 64.09]
Statistical Analysis 35: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 13]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 43.16, 95% CI 2-sided [29.56 to 56.75]
Statistical Analysis 36: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 13]; Test type: Superiority or Other; p = 0.087, Cochran-Mantel-Haenszel; CMH adjusted proportions = 7.91, 95% CI 2-sided [-1.15 to 16.97]
Statistical Analysis 37: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 16, analysis 19]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 58.12, 95% CI 2-sided [45.24 to 71.00]
Statistical Analysis 38: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 19]; Test type: Superiority or Other; p = 0.071, Cochran-Mantel-Haenszel; CMH adjusted proportions = 7.23, 95% CI 2-sided [-0.63 to 15.10]
Statistical Analysis 39: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 19]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 15.12, 95% CI 2-sided [6.55 to 23.69]
Statistical Analysis 40: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 19]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 50.74, 95% CI 2-sided [37.39 to 64.09]
Statistical Analysis 41: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 19]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 43.16, 95% CI 2-sided [29.56 to 56.75]
Statistical Analysis 42: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 19]; Test type: Superiority or Other; p = 0.087, Cochran-Mantel-Haenszel; CMH adjusted proportions = 7.91, 95% CI 2-sided [-1.15 to 16.97]
Statistical Analysis 43: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 16, analysis 25]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 58.12, 95% CI 2-sided [45.24 to 71.00]
Statistical Analysis 44: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 25]; Test type: Superiority or Other; p = 0.071, Cochran-Mantel-Haenszel; CMH adjusted proportions = 7.23, 95% CI 2-sided [-0.63 to 15.10]
Statistical Analysis 45: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 25]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 15.12, 95% CI 2-sided [6.55 to 23.69]
Statistical Analysis 46: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 25]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 50.74, 95% CI 2-sided [37.39 to 64.09]
Statistical Analysis 47: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 25]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 43.16, 95% CI 2-sided [29.56 to 56.75]
Statistical Analysis 48: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 25]; Test type: Superiority or Other; p = 0.087, Cochran-Mantel-Haenszel; CMH adjusted proportions = 7.91, 95% CI 2-sided [-1.15 to 16.97]
Statistical Analysis 49: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 16, analysis 31]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 58.12, 95% CI 2-sided [45.24 to 71.00]
Statistical Analysis 50: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 31]; Test type: Superiority or Other; p = 0.071, Cochran-Mantel-Haenszel; CMH adjusted proportions = 7.23, 95% CI 2-sided [-0.63 to 15.10]
Statistical Analysis 51: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 31]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 15.12, 95% CI 2-sided [6.55 to 23.69]
Statistical Analysis 52: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 31]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 50.74, 95% CI 2-sided [37.39 to 64.09]
Statistical Analysis 53: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 31]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 43.16, 95% CI 2-sided [29.56 to 56.75]
Statistical Analysis 54: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 31]; Test type: Superiority or Other; p = 0.087, Cochran-Mantel-Haenszel; CMH adjusted proportions = 7.91, 95% CI 2-sided [-1.15 to 16.97]
Statistical Analysis 55: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 16, analysis 37]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 58.12, 95% CI 2-sided [45.24 to 71.00]
Statistical Analysis 56: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 37]; Test type: Superiority or Other; p = 0.071, Cochran-Mantel-Haenszel; CMH adjusted proportions = 7.23, 95% CI 2-sided [-0.63 to 15.10]
Statistical Analysis 57: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 37]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 15.12, 95% CI 2-sided [6.55 to 23.69]
Statistical Analysis 58: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 37]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 50.74, 95% CI 2-sided [37.39 to 64.09]
Statistical Analysis 59: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 37]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 43.16, 95% CI 2-sided [29.56 to 56.75]
Statistical Analysis 60: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 37]; Test type: Superiority or Other; p = 0.087, Cochran-Mantel-Haenszel; CMH adjusted proportions = 7.91, 95% CI 2-sided [-1.15 to 16.97]
Statistical Analysis 61: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 16, analysis 43]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 58.12, 95% CI 2-sided [45.24 to 71.00]
Statistical Analysis 62: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 43]; Test type: Superiority or Other; p = 0.071, Cochran-Mantel-Haenszel; CMH adjusted proportions = 7.23, 95% CI 2-sided [-0.63 to 15.10]
Statistical Analysis 63: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 43]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 15.12, 95% CI 2-sided [6.55 to 23.69]
Statistical Analysis 64: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 43]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 50.74, 95% CI [37.39 to 64.09]
Statistical Analysis 65: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 43]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 43.16, 95% CI [29.56 to 56.75]
Statistical Analysis 66: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 43]; Test type: Superiority or Other; p = 0.087, Cochran-Mantel-Haenszel; CMH adjusted proportions = 7.91, 95% CI [-1.15 to 16.97]
Statistical Analysis 67: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 16, analysis 49]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 58.12, 95% CI [45.24 to 71.00]
Statistical Analysis 68: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 49]; Test type: Superiority or Other; p = 0.071, Cochran-Mantel-Haenszel; CMH adjusted proportions = 7.23, 95% CI [-0.63 to 15.10]
Statistical Analysis 69: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 49]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 15.12, 95% CI [6.55 to 23.69]
Statistical Analysis 70: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 49]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 50.74, 95% CI 2-sided [37.39 to 64.09]
Statistical Analysis 71: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 49]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 43.16, 95% CI 2-sided [29.56 to 56.75]
Statistical Analysis 72: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 49]; Test type: Superiority or Other; p = 0.087, Cochran-Mantel-Haenszel; CMH adjusted proportions = 7.91, 95% CI [-1.15 to 16.97]
Statistical Analysis 73: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 16, analysis 55]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 58.12, 95% CI 2-sided [45.24 to 71.00]
Statistical Analysis 74: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 55]; Test type: Superiority or Other; p = 0.071, Cochran-Mantel-Haenszel; CMH adjusted proportions = 7.23, 95% CI [-0.63 to 15.10]
Statistical Analysis 75: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 55]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 15.12, 95% CI 2-sided [6.55 to 23.69]
Statistical Analysis 76: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 55]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 50.74, 95% CI 2-sided [37.39 to 64.09]
Statistical Analysis 77: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 55]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 43.16, 95% CI [29.56 to 56.75]
Statistical Analysis 78: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 55]; Test type: Superiority or Other; p = 0.087, Cochran-Mantel-Haenszel; CMH adjusted proportions = 7.91, 95% CI 2-sided [-1.15 to 16.97]
Statistical Analysis 79: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 16, analysis 61]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 58.12, 95% CI 2-sided [45.24 to 71.00]
Statistical Analysis 80: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 61]; Test type: Superiority or Other; p = 0.071, Cochran-Mantel-Haenszel; CMH adjusted proportions = 7.23, 95% CI [-0.63 to 15.10]
Statistical Analysis 81: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 61]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 15.12, 95% CI [6.55 to 23.69]
Statistical Analysis 82: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 61]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 50.74, 95% CI [37.39 to 64.09]
Statistical Analysis 83: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 61]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 43.16, 95% CI 2-sided [29.56 to 56.75]
Statistical Analysis 84: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 61]; Test type: Superiority or Other; p = 0.087, Cochran-Mantel-Haenszel; CMH adjusted proportions = 7.91, 95% CI 2-sided [-1.15 to 16.97]
Statistical Analysis 85: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 16, analysis 67]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 58.12, 95% CI 2-sided [45.24 to 71.00]
Statistical Analysis 86: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 67]; Test type: Superiority or Other; p = 0.071, Cochran-Mantel-Haenszel; CMH adjusted proportions = 7.23, 95% CI 2-sided [-0.63 to 15.10]
Statistical Analysis 87: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 67]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 15.12, 95% CI 2-sided [6.55 to 23.69]
Statistical Analysis 88: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 67]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 50.74, 95% CI 2-sided [37.39 to 64.09]
Statistical Analysis 89: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 67]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 43.16, 95% CI 2-sided [29.56 to 56.75]
Statistical Analysis 90: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 67]; Test type: Superiority or Other; p = 0.087, Cochran-Mantel-Haenszel; CMH adjusted proportions = 7.91, 95% CI 2-sided [-1.15 to 16.97]

18. Other Pre Specified Outcome: Cumulative Percentage of Participants With Meaningful Relief
Description: Percentage of participants with meaningful relief was reported. Participants evaluated time to meaningful relief by stopping a second stopwatch labeled "meaningful relief" at the moment they first began to experience meaningful relief. Stopwatch was active up to 12 hours after dosing or until stopped by participant, or participant became treatment failure prior to depressing the second stopwatch. Treatment failure was defined as participant taking rescue medication, or discontinuing due to lack of efficacy.
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 hours post-dose
Population: FAS included all randomized participants who were dosed with the study medication and provided a baseline assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ibuprofen 250 mg + Acetaminophen 500 mg | Ibuprofen 250 mg | Acetaminophen 650 mg
Number analyzed (Participants) | 56 | 172 | 175 | 165
percentage of participants
  0.25 hour | 0.0 | 1.2 | 0.0 | 1.8
  0.5 hour | 0.0 | 21.5 | 13.7 | 21.8
  1 hour | 3.6 | 59.3 | 46.3 | 52.1
  1.5 hour | 8.9 | 68.6 | 60.0 | 58.2
  2 hour | 16.1 | 82.0 | 75.4 | 67.3
  3 hour | 21.4 | 82.0 | 75.4 | 67.3
  4 hour | 23.2 | 83.1 | 77.1 | 67.9
  5 hour | 26.8 | 84.3 | 78.3 | 69.1
  6 hour | 26.8 | 85.5 | 78.9 | 69.7
  7 hour | 26.8 | 85.5 | 78.9 | 69.7
  8 hour | 26.8 | 85.5 | 78.9 | 70.3
  9 hour | 26.8 | 85.5 | 78.9 | 71.5
  10 hour | 28.6 | 85.5 | 79.4 | 71.5
  11 hour | 28.6 | 85.5 | 79.4 | 71.5
  12 hour | 28.6 | 85.5 | 79.4 | 71.5
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; p = 0.156, Cochran-Mantel-Haenszel; CMH adjusted proportions = 1.16, 95% CI 2-sided [-0.44 to 2.75]
Statistical Analysis 2: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; p = 0.155, Cochran-Mantel-Haenszel; CMH adjusted proportions = 1.16, 95% CI 2-sided [-0.44 to 2.76]
Statistical Analysis 3: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; p = 0.605, Cochran-Mantel-Haenszel; CMH adjusted proportions = -0.68, 95% CI 2-sided [-3.27 to 1.90]
Statistical Analysis 4: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; p = 0.079, Cochran-Mantel-Haenszel; CMH adjusted proportions = 1.84, 95% CI 2-sided [-0.21 to 3.89]
Statistical Analysis 5: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; p = 0.078, Cochran-Mantel-Haenszel; CMH adjusted proportions = -1.85, 95% CI 2-sided [-3.90 to 0.21]
Statistical Analysis 6: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 17, analysis 7]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 21.47, 95% CI 2-sided [15.33 to 27.62]
Statistical Analysis 7: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 17, analysis 7]; Test type: Superiority or Other; p = 0.056, Cochran-Mantel-Haenszel; Cumulative Percentage of Participants wi = 7.79, 95% CI 2-sided [-0.19 to 15.77]
Statistical Analysis 8: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 17, analysis 7]; Test type: Superiority or Other; p = 0.934, Cochran-Mantel-Haenszel; CMH adjusted proportions = -0.37, 95% CI 2-sided [-9.18 to 8.43]
Statistical Analysis 9: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 17, analysis 7]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 13.67, 95% CI 2-sided [8.58 to 18.77]
Statistical Analysis 10: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 17, analysis 7]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 21.96, 95% CI 2-sided [15.64 to 28.28]
Statistical Analysis 11: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 17, analysis 7]; Test type: Superiority or Other; p = 0.050, Cochran-Mantel-Haenszel; CMH adjusted proportions = -8.21, 95% CI 2-sided [-16.40 to -0.01]
Statistical Analysis 12: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 17, analysis 13]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 55.89, 95% CI 2-sided [47.05 to 64.73]
Statistical Analysis 13: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 17, analysis 13]; Test type: Superiority or Other; p = 0.015, Cochran-Mantel-Haenszel; CMH adjusted proportions = 12.99, 95% CI 2-sided [2.50 to 23.49]
Statistical Analysis 14: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 17, analysis 13]; Test type: Superiority or Other; p = 0.188, Cochran-Mantel-Haenszel; CMH adjusted proportions = 7.16, 95% CI 2-sided [-3.51 to 17.82]
Statistical Analysis 15: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 17, analysis 13]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 42.61, 95% CI 2-sided [33.85 to 51.38]
Statistical Analysis 16: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 17, analysis 13]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 48.58, 95% CI 2-sided [39.63 to 57.54]
Statistical Analysis 17: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 17, analysis 13]; Test type: Superiority or Other; p = 0.266, Cochran-Mantel-Haenszel; CMH adjusted proportions = -5.98, 95% CI 2-sided [-16.51 to 4.55]
Statistical Analysis 18: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 59.77, 95% CI 2-sided [49.63 to 69.90]
Statistical Analysis 19: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; p = 0.094, Cochran-Mantel-Haenszel; CMH adjusted proportions = 8.62, 95% CI 2-sided [-1.46 to 18.69]
Statistical Analysis 20: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; p = 0.047, Cochran-Mantel-Haenszel; CMH adjusted proportions = 10.43, 95% CI 2-sided [0.15 to 20.72]
Statistical Analysis 21: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 50.95, 95% CI 2-sided [40.50 to 61.40]
Statistical Analysis 22: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 49.34, 95% CI 2-sided [38.79 to 59.89]
Statistical Analysis 23: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; p = 0.734, Cochran-Mantel-Haenszel; CMH adjusted proportions = 1.79, 95% CI 2-sided [-8.56 to 12.14]
Statistical Analysis 24: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 16, analysis 7]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 58.46, 95% CI 2-sided [46.88 to 70.03]
Statistical Analysis 25: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 7]; Test type: Superiority or Other; p = 0.152, Cochran-Mantel-Haenszel; CMH adjusted proportions = 7.01, 95% CI 2-sided [-2.57 to 16.59]
Statistical Analysis 26: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 7]; Test type: Superiority or Other; p = 0.073, Cochran-Mantel-Haenszel; CMH adjusted proportions = 9.00, 95% CI 2-sided [-0.83 to 19.82]
Statistical Analysis 27: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 7]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 51.30, 95% CI 2-sided [39.38 to 63.21]
Statistical Analysis 28: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 7]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 49.49, 95% CI 2-sided [37.50 to 61.47]
Statistical Analysis 29: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 7]; Test type: Superiority or Other; p = 0.694, Cochran-Mantel-Haenszel; CMH adjusted proportions = 1.99, 95% CI 2-sided [-7.91 to 11.89]
Statistical Analysis 30: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 16, analysis 13]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 60.61, 95% CI 2-sided [48.37 to 72.84]
Statistical Analysis 31: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 13]; Test type: Superiority or Other; p = 0.135, Cochran-Mantel-Haenszel; CMH adjusted proportions = 6.58, 95% CI 2-sided [-2.05 to 15.20]
Statistical Analysis 32: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 13]; Test type: Superiority or Other; p = 0.002, Cochran-Mantel-Haenszel; CMH adjusted proportions = 14.74, 95% CI 2-sided [5.50 to 23.97]
Statistical Analysis 33: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 13]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 53.82, 95% CI 2-sided [41.31 to 66.32]
Statistical Analysis 34: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 13]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 45.93, 95% CI 2-sided [33.21 to 58.66]
Statistical Analysis 35: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 13]; Test type: Superiority or Other; p = 0.091, Cochran-Mantel-Haenszel; CMH adjusted proportions = 8.18, 95% CI 2-sided [-1.32 to 17.69]
Statistical Analysis 36: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 16, analysis 19]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 60.00, 95% CI 2-sided [47.59 to 72.42]
Statistical Analysis 37: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 19]; Test type: Superiority or Other; p = 0.159, Cochran-Mantel-Haenszel; CMH adjusted proportions = 6.03, 95% CI 2-sided [-2.36 to 14.43]
Statistical Analysis 38: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 19]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 15.32, 95% CI 2-sided [6.23 to 24.41]
Statistical Analysis 39: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 19]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 53.79, 95% CI 2-sided [41.08 to 66.50]
Statistical Analysis 40: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 19]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 44.76, 95% CI 2-sided [31.72 to 57.81]
Statistical Analysis 41: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 19]; Test type: Superiority or Other; p = 0.052, Cochran-Mantel-Haenszel; CMH adjusted proportions = 9.28, 95% CI 2-sided [-0.08 to 18.64]
Statistical Analysis 42: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 16, analysis 25]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 57.57, 95% CI 2-sided [44.75 to 70.39]
Statistical Analysis 43: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 25]; Test type: Superiority or Other; p = 0.147, Cochran-Mantel-Haenszel; CMH adjusted proportions = 6.06, 95% CI 2-sided [-2.13 to 14.25]
Statistical Analysis 44: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 25]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 15.30, 95% CI 2-sided [6.39 to 24.21]
Statistical Analysis 45: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 25]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 51.32, 95% CI 2-sided [38.16 to 64.48]
Statistical Analysis 46: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 25]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 42.28, 95% CI 2-sided [28.74 to 55.82]
Statistical Analysis 47: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 25]; Test type: Superiority or Other; p = 0.049, Cochran-Mantel-Haenszel; CMH adjusted proportions = 9.27, 95% CI 2-sided [0.04 to 18.49]
Statistical Analysis 48: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 16, analysis 31]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 58.71, 95% CI 2-sided [45.93 to 71.49]
Statistical Analysis 49: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 31]; Test type: Superiority or Other; p = 0.105, Cochran-Mantel-Haenszel; CMH adjusted proportions = 6.64, 95% CI 2-sided [-1.38 to 14.67]
Statistical Analysis 50: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 31]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 15.86, 95% CI 2-sided [7.08 to 24.63]
Statistical Analysis 51: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 31]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 51.90, 95% CI 2-sided [38.76 to 65.04]
Statistical Analysis 52: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 31]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 42.94, 95% CI 2-sided [29.44 to 56.44]
Statistical Analysis 53: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 31]; Test type: Superiority or Other; p = 0.048, Cochran-Mantel-Haenszel; CMH adjusted proportions = 9.23, 95% CI 2-sided [0.06 to 18.40]
Statistical Analysis 54: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 16, analysis 37]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 58.71, 95% CI 2-sided [45.93 to 71.49]
Statistical Analysis 55: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 37]; Test type: Superiority or Other; p = 0.105, Cochran-Mantel-Haenszel; CMH adjusted proportions = 6.64, 95% CI 2-sided [-1.38 to 14.67]
Statistical Analysis 56: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 37]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 15.86, 95% CI 2-sided [7.08 to 24.63]
Statistical Analysis 57: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 37]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 51.90, 95% CI 2-sided [38.76 to 65.04]
Statistical Analysis 58: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 37]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 42.94, 95% CI 2-sided [29.44 to 56.44]
Statistical Analysis 59: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 37]; Test type: Superiority or Other; p = 0.048, Cochran-Mantel-Haenszel; CMH adjusted proportions = 9.23, 95% CI 2-sided [0.06 to 18.40]
Statistical Analysis 60: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 16, analysis 43]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 58.71, 95% CI [45.93 to 71.49]
Statistical Analysis 61: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 43]; Test type: Superiority or Other; p = 0.105, Cochran-Mantel-Haenszel; CMH adjusted proportions = 6.64, 95% CI 2-sided [-1.38 to 14.67]
Statistical Analysis 62: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 43]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 15.23, 95% CI 2-sided [6.48 to 23.97]
Statistical Analysis 63: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 43]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 51.90, 95% CI [38.76 to 65.04]
Statistical Analysis 64: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 43]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 43.61, 95% CI 2-sided [30.15 to 57.07]
Statistical Analysis 65: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 43]; Test type: Superiority or Other; p = 0.065, Cochran-Mantel-Haenszel; CMH adjusted proportions = 8.61, 95% CI 2-sided [-0.55 to 17.76]
Statistical Analysis 66: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 16, analysis 49]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 58.71, 95% CI [45.93 to 71.49]
Statistical Analysis 67: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 49]; Test type: Superiority or Other; p = 0.105, Cochran-Mantel-Haenszel; CMH adjusted proportions = 6.64, 95% CI 2-sided [-1.38 to 14.67]
Statistical Analysis 68: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 49]; Test type: Superiority or Other; p = 0.002, Cochran-Mantel-Haenszel; CMH adjusted proportions = 13.98, 95% CI 2-sided [5.30 to 22.67]
Statistical Analysis 69: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 49]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 51.90, 95% CI 2-sided [38.76 to 65.04]
Statistical Analysis 70: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 49]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 44.89, 95% CI [31.51 to 58.26]
Statistical Analysis 71: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 49]; Test type: Superiority or Other; p = 0.113, Cochran-Mantel-Haenszel; CMH adjusted proportions = 7.36, 95% CI 2-sided [-1.73 to 16.45]
Statistical Analysis 72: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 16, analysis 55]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 56.94, 95% CI 2-sided [43.95 to 69.94]
Statistical Analysis 73: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 55]; Test type: Superiority or Other; p = 0.136, Cochran-Mantel-Haenszel; CMH adjusted proportions = 6.07, 95% CI 2-sided [-1.91 to 14.05]
Statistical Analysis 74: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 55]; Test type: Superiority or Other; p = 0.002, Cochran-Mantel-Haenszel; CMH adjusted proportions = 13.98, 95% CI 2-sided [5.30 to 22.67]
Statistical Analysis 75: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 55]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 50.74, 95% CI 2-sided [37.39 to 64.09]
Statistical Analysis 76: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 55]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 43.16, 95% CI 2-sided [29.56 to 56.75]
Statistical Analysis 77: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 55]; Test type: Superiority or Other; p = 0.087, Cochran-Mantel-Haenszel; CMH adjusted proportions = 7.91, 95% CI 2-sided [-1.15 to 16.97]
Statistical Analysis 78: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 16, analysis 61]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 56.94, 95% CI 2-sided [43.95 to 69.94]
Statistical Analysis 79: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 61]; Test type: Superiority or Other; p = 0.136, Cochran-Mantel-Haenszel; CMH adjusted proportions = 6.07, 95% CI 2-sided [-1.91 to 14.05]
Statistical Analysis 80: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 61]; Test type: Superiority or Other; p = 0.002, Cochran-Mantel-Haenszel; CMH adjusted proportions = 13.98, 95% CI 2-sided [5.30 to 22.67]
Statistical Analysis 81: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 61]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 50.74, 95% CI 2-sided [37.39 to 64.09]
Statistical Analysis 82: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 61]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 43.16, 95% CI 2-sided [29.56 to 56.75]
Statistical Analysis 83: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 61]; Test type: Superiority or Other; p = 0.087, Cochran-Mantel-Haenszel; CMH adjusted proportions = 7.91, 95% CI 2-sided [-1.15 to 16.97]
Statistical Analysis 84: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 16, analysis 67]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 56.94, 95% CI 2-sided [43.95 to 69.94]
Statistical Analysis 85: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 67]; Test type: Superiority or Other; p = 0.136, Cochran-Mantel-Haenszel; CMH adjusted proportions = 6.07, 95% CI 2-sided [-1.91 to 14.05]
Statistical Analysis 86: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 67]; Test type: Superiority or Other; p = 0.002, Cochran-Mantel-Haenszel; CMH adjusted proportions = 13.98, 95% CI 2-sided [5.30 to 22.67]
Statistical Analysis 87: Comparison: Placebo vs Ibuprofen 250 mg; [analysis description as in outcome 16, analysis 67]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 50.74, 95% CI 2-sided [37.39 to 64.09]
Statistical Analysis 88: Comparison: Placebo vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 67]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH adjusted proportions = 43.16, 95% CI 2-sided [29.56 to 56.75]
Statistical Analysis 89: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; [analysis description as in outcome 16, analysis 67]; Test type: Superiority or Other; p = 0.087, Cochran-Mantel-Haenszel; CMH adjusted proportions = 7.91, 95% CI 2-sided [-1.15 to 16.97]

19. Other Pre Specified Outcome: Participant's Global Evaluation of Study Medication
Description: Participant global evaluation of study medication was performed at the 12-hour time point or immediately before taking the rescue medication. It was scored on a 6-point categorical scale where 0= Very poor, 1= Poor, 2= Fair, 3= Good, 4= Very Good and 5= Excellent.
Time Frame: 0 to 12 hours post-dose
Population: FAS included all randomized participants who were dosed with the study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen 250 mg + Acetaminophen 500 mg | Ibuprofen 250 mg | Acetaminophen 650 mg
Number analyzed (Participants) | 56 | 172 | 175 | 165
units on a scale | 1.0 (1.4) | 3.4 (1.2) | 3.0 (1.4) | 2.6 (1.5)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; p-value was calculated from CMH test with modified ridit scores, controlling for baseline categorical PSR and gender; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 250 mg; p-value was calculated from CMH test with modified ridit scores, controlling for baseline categorical PSR and gender; Test type: Superiority or Other; p = 0.004, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Acetaminophen 650 mg; p-value was calculated from CMH test with modified ridit scores, controlling for baseline categorical PSR and gender; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen 250 mg; p-value was calculated from CMH test with modified ridit scores, controlling for baseline categorical PSR and gender; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Placebo vs Acetaminophen 650 mg; p-value was calculated from CMH test with modified ridit scores, controlling for baseline categorical PSR and gender; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Ibuprofen 250 mg vs Acetaminophen 650 mg; p-value was calculated from CMH test with modified ridit scores, controlling for baseline categorical PSR and gender; Test type: Superiority or Other; p = 0.003, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Arm/Group | Placebo | Ibuprofen 250 mg + Acetaminophen 500 mg | Ibuprofen 250 mg | Acetaminophen 650 mg
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/172 | 0/175 | 0/165
Other Adverse Events (participants affected / at risk) | 19/56 | 21/172 | 37/175 | 41/165
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=56) | Ibuprofen 250 mg + Acetaminophen 500 mg (N=172) | Ibuprofen 250 mg (N=175) | Acetaminophen 650 mg (N=165)
Nausea (Gastrointestinal disorders) | 17 | 17 | 24 | 33
Vomiting (Gastrointestinal disorders) | 11 | 7 | 15 | 20
Dizziness (Nervous system disorders) | 4 | 5 | 6 | 12
Headache (Nervous system disorders) | 0 | 0 | 3 | 4
Flushing (Vascular disorders) | 2 | 0 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.